CLINICAL TRIAL: NCT00880893
Title: Immunogenicity and Large-Scale Safety of Tetravalent Dengue Vaccine in Healthy Subjects Aged 2 to 45 Years in Singapore
Brief Title: Study of Sanofi Pasteur's CYD Dengue Vaccine in Healthy Subjects in Singapore
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CYD28; 2014-001713-26 (EudraCT Number)
Record Dates: First submitted 2009-04-13; First posted 2009-04-14 (Estimated); Results first posted 2019-07-29 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Dengue Fever; Dengue Hemorrhagic Fever; Dengue Virus; Dengue Diseases
Keywords: Dengue virus; Dengue fever; Dengue Hemorrhagic fever; Dengue diseases; Sanofi Pasteur's CYD Dengue Vaccine
MeSH Terms: conditions — Dengue; Severe Dengue | interventions — Hepatitis A Vaccines; Sodium Chloride; vaxigrip

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: An observer-design for the first vaccination and a single-blind design for the second and third vaccination were chosen to minimize the bias of the vaccine evaluation. The Investigator in charge of safety evaluation, the Sponsor, and the participants/parents did not know which vaccine was administrated at the first visit. For the second and third vaccinations, the participants/parents did not know which vaccine was administered.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CYD Dengue Vaccine Group (Experimental): Participant's received the CYD Dengue Vaccine at 0, 6, and 12 months as first, second, and third vaccinations, respectively.
  Interventions: Biological: CYD Dengue vaccine
- Placebo Group (Sham Comparator): All participants received a placebo at first vaccination (Month 0). Participants <12 years received hepatitis A at second (Month 6) and third (Month 12) vaccinations. Participants >= 12 years received influenza vaccine of Northern and Southern hemisphere formulations at second (Month 6) and third (Month 12) vaccinations.
  Interventions: Biological: NaCl + influenza virus or hepatitis A vaccine

INTERVENTIONS:
Biological: CYD Dengue vaccine — 0.5 mL, Subcutaneous on Day 0, Months 6 and 12
  Other Names: Sanofi Pasteur's CYD Dengue Vaccine
  Arms: CYD Dengue Vaccine Group
Biological: NaCl + influenza virus or hepatitis A vaccine — 0.5 mL, Subcutaneous (Intramuscular - Hepatitis A)
  Other Names: NaCl 0.9%; Vaxigrip®; Havrix® pediatric formulation
  Arms: Placebo Group

SUMMARY:
Primary Objectives:

* To evaluate safety after each CYD Dengue vaccination in terms of injection site and systemic reactogenicity.
* To evaluate the occurrence of Serious Adverse Events (SAEs) throughout the trial period.
* To evaluate the humoral immune response to each CYD Dengue serotype after each vaccination in a subset of participants.

Secondary Objectives:

* To evaluate the persistence of the humoral immune response during 4 years after the last vaccination in a subset of participants.

DETAILED DESCRIPTION:
This was a multicenter trial involving three vaccinations one each at 0, 6 and 12 months over a period of 1 year, and a 4-year follow-up following the last vaccination.

ELIGIBILITY:
Inclusion Criteria :

* Aged from 2 to 45 years on the day of inclusion.
* Participant in good health, based on medical history and physical examination.
* Provision of informed consent form (and assent form for participants aged 6 to 12 years) signed by the participant and by the parent(s) or another legally acceptable representative for participants aged less than 21 years.
* Participants and parent(s)/legally acceptable representative able to attend all scheduled visits and comply with all trial procedures.
* For a woman of child-bearing potential, avoid becoming pregnant (use of an effective method of contraception or abstinence) for at least 4 weeks before the first vaccination until 4 weeks after the last vaccination.

Exclusion Criteria :

* Febrile illness (temperature >= 37.5°C) or moderate or severe acute illness/infection on the day of the first vaccination, according to Investigator judgment.
* For a woman of child-bearing potential, known pregnancy or positive urine pregnancy test on the day of inclusion.
* Breast-feeding woman.
* Known systemic hypersensitivity to any of the components of the trial vaccines (especially egg proteins or neomycin) or history of a life-threatening reaction to the trial vaccines or to a vaccine containing any of the same substances.
* Personal or family history of thymic pathology or myasthenia.
* Previous hepatitis A vaccination (for children only).
* Known or suspected congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the past 6 months, or long-term systemic corticosteroid therapy.
* Chronic illness at a stage that could interfere with trial conduct or completion, in the opinion of the Investigator.
* Receipt of blood or blood-derived products in the past 3 months that might interfere with the assessment of immune response.
* Participation in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure in the 4 weeks preceding the first trial vaccination.
* Planned participation in another clinical trial during the 18 coming months.
* Receipt of any vaccine in the 4 weeks preceding the first trial vaccination.
* Planned receipt of any vaccine in the 4 weeks following the first trial vaccination.
* Participant deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized without his/her consent.
* Current or past alcohol abuse or drug addiction that may interfere with the participants ability to comply with trial procedures.
* Participant who plans to move to another country within the 18 coming months.

Ages: 2 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1198 (Actual)
Dates: Start 2009-04-07 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2014-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (1):
- Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Result] Harenberg A, Begue S, Mamessier A, Gimenez-Fourage S, Ching Seah C, Wei Liang A, Li Ng J, Yun Toh X, Archuleta S, Wilder-Smith A, Shek LP, Wartel-Tram A, Bouckenooghe A, Lang J, Crevat D, Caillet C, Guy B. Persistence of Th1/Tc1 responses one year after tetravalent dengue vaccination in adults and adolescents in Singapore. Hum Vaccin Immunother. 2013 Nov;9(11):2317-25. doi: 10.4161/hv.25562. Epub 2013 Jul 9. PMID 23839107
- [Derived] Leo YS, Wilder-Smith A, Archuleta S, Shek LP, Chong CY, Leong HN, Low CY, Oh ML, Bouckenooghe A, Wartel TA, Crevat D. Immunogenicity and safety of recombinant tetravalent dengue vaccine (CYD-TDV) in individuals aged 2-45 y: Phase II randomized controlled trial in Singapore. Hum Vaccin Immunother. 2012 Sep;8(9):1259-71. doi: 10.4161/hv.21224. Epub 2012 Aug 16. PMID 22894958
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled from 07 April 2009 to 08 October 2009 at 5 clinical sites in Singapore.
Pre-assignment Details: A total of 1198 participants who met all of the inclusion criteria and none of the exclusion criteria were enrolled and randomized.
Groups:
- CYD Dengue Vaccine Group: Participants received the CYD dengue vaccine at 0, 6, and 12 months as first, second, and third vaccinations, respectively.
- Placebo Group: All participants received a placebo at first vaccination (Month 0). Participants <12 years received hepatitis A at second (Month 6) and third (Month 12) vaccinations. Participants >=12 years received influenza vaccine of Northern and Southern hemisphere formulations at second (Month 6) and third (Month 12) vaccinations.
Period: Overall Study
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Started | 898 | 300
Completed | 791 | 255
Not Completed | 107 | 45
Not completed — Protocol Violation | 13 | 1
Not completed — Withdrawal by Subject | 15 | 11
Not completed — Lost to Follow-up | 76 | 33
Not completed — Serious adverse event | 3 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on Safety analysis set which included all participants who had received at least one dose of CYD dengue or control vaccine.
Groups:
- Total: Total of all reporting groups
Arm/Group | CYD Dengue Vaccine Group | Placebo Group | Total
Number analyzed (Participants) | 898 | 300 | 1198
Age, Continuous [Mean (Standard Deviation); unit: Years] | 22.1 (12.0) | 21.7 (11.8) | 22.0 (11.9)
Age, Customized [Count of Participants; unit: Participants]
  2-11 years | 236 | 80 | 316
  12-17 years | 141 | 46 | 187
  18-45 years | 521 | 174 | 695
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 471 | 139 | 610
  Male | 427 | 161 | 588

OUTCOME MEASURES:

1. Primary Outcome: Percentage of All Participants Reporting Solicited Injection-site and Systemic Reactions Following Each Injection With CYD Dengue Vaccine or Placebo
Description: Solicited injection site reactions: Pain, Erythema, and Swelling. Solicited systemic reactions: Fever, Headache, Malaise, Myalgia, and Asthenia. Grade 3 Solicited injection site reactions (2-11 years): Pain, incapacitating, unable to perform usual activities; Erythema and Swelling, >=5 cm. Grade 3 Solicited injection site reactions (adolescents and adults: >=12 years): Pain, significant; prevents daily activity; Erythema and Swelling: >10 cm. Grade 3 Solicited systemic reactions (all participants): Fever, >=39.0°C; Headache, Malaise, Myalgia, and Asthenia: significant; prevents daily activity.
Time Frame: Day 0 up to 14 days post-any and each injection
Population: Analysis was performed on Safety analysis set. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 898 | 300
Percentage of participants
  Injection site Pain; Post-Any Injection: number analyzed (Participants) | 892 | 297
  Injection site Pain; Post-Any Injection | 53.9 | 66.7
  Grade 3 Injection site Pain; Post-Any Injection: number analyzed (Participants) | 892 | 297
  Grade 3 Injection site Pain; Post-Any Injection | 1.0 | 2.0
  Injection site Erythema; Post-Any Injection: number analyzed (Participants) | 891 | 297
  Injection site Erythema; Post-Any Injection | 7.2 | 15.2
  Grade 3 Inj. site Erythema; Post-Any Inj.: number analyzed (Participants) | 891 | 297
  Grade 3 Inj. site Erythema; Post-Any Inj. | 0.0 | 0.0
  Injection site Swelling; Post-Any Injection: number analyzed (Participants) | 892 | 297
  Injection site Swelling; Post-Any Injection | 4.1 | 8.4
  Grade 3 Inj. site Swelling; Post-Any Inj.: number analyzed (Participants) | 892 | 297
  Grade 3 Inj. site Swelling; Post-Any Inj. | 0.0 | 0.0
  Injection site Pain; Post-Injection 1: number analyzed (Participants) | 892 | 297
  Injection site Pain; Post-Injection 1 | 31.3 | 21.9
  Grade 3 Injection site Pain; Post- Injection 1: number analyzed (Participants) | 892 | 297
  Grade 3 Injection site Pain; Post- Injection 1 | 0.3 | 0.7
  Injection site Erythema; Post-Injection 1: number analyzed (Participants) | 891 | 297
  Injection site Erythema; Post-Injection 1 | 2.0 | 2.0
  Grade 3 Injection site Erythema; Post- Injection 1: number analyzed (Participants) | 891 | 297
  Grade 3 Injection site Erythema; Post- Injection 1 | 0.0 | 0.0
  Injection site Swelling; Post-Injection 1: number analyzed (Participants) | 892 | 297
  Injection site Swelling; Post-Injection 1 | 1.1 | 1.7
  Grade 3 Injection site Swelling; Post- Injection 1: number analyzed (Participants) | 892 | 297
  Grade 3 Injection site Swelling; Post- Injection 1 | 0.0 | 0.0
  Injection site Pain; Post-Injection 2: number analyzed (Participants) | 859 | 285
  Injection site Pain; Post-Injection 2 | 36.9 | 54.4
  Grade 3 Injection site Pain; Post- Injection 2: number analyzed (Participants) | 859 | 285
  Grade 3 Injection site Pain; Post- Injection 2 | 0.5 | 0.7
  Injection site Erythema; Post-Injection 2: number analyzed (Participants) | 859 | 285
  Injection site Erythema; Post-Injection 2 | 3.4 | 8.8
  Grade 3 Injection site Erythema; Post- Injection 2: number analyzed (Participants) | 859 | 285
  Grade 3 Injection site Erythema; Post- Injection 2 | 0.0 | 0.0
  Injection site Swelling; Post-Injection 2: number analyzed (Participants) | 859 | 285
  Injection site Swelling; Post-Injection 2 | 1.4 | 3.5
  Grade 3 Injection site Swelling; Post- Injection 2: number analyzed (Participants) | 859 | 285
  Grade 3 Injection site Swelling; Post- Injection 2 | 0.0 | 0.0
  Injection site Pain; Post-Injection 3: number analyzed (Participants) | 836 | 278
  Injection site Pain; Post-Injection 3 | 34.9 | 50.0
  Grade 3 Injection site Pain; Post- Injection 3: number analyzed (Participants) | 836 | 278
  Grade 3 Injection site Pain; Post- Injection 3 | 0.2 | 0.7
  Injection site Erythema; Post-Injection 3: number analyzed (Participants) | 836 | 278
  Injection site Erythema; Post-Injection 3 | 3.8 | 9.4
  Grade 3 Injection site Erythema; Post- Injection 3: number analyzed (Participants) | 836 | 278
  Grade 3 Injection site Erythema; Post- Injection 3 | 0.0 | 0.0
  Injection site Swelling; Post-Injection 3: number analyzed (Participants) | 836 | 278
  Injection site Swelling; Post-Injection 3 | 2.6 | 5.8
  Grade 3 Injection site Swelling; Post- Injection 3: number analyzed (Participants) | 836 | 278
  Grade 3 Injection site Swelling; Post- Injection 3 | 0.0 | 0.0
  Fever; Post-Any Injection: number analyzed (Participants) | 892 | 297
  Fever; Post-Any Injection | 11.3 | 7.4
  Grade 3 Fever; Post-Any Injection: number analyzed (Participants) | 892 | 297
  Grade 3 Fever; Post-Any Injection | 1.9 | 1.0
  Headache; Post-Any Injection: number analyzed (Participants) | 891 | 297
  Headache; Post-Any Injection | 45.1 | 38.4
  Grade 3 Headache; Post-Any Injection: number analyzed (Participants) | 891 | 297
  Grade 3 Headache; Post-Any Injection | 3.8 | 2.7
  Malaise; Post-Any Injection: number analyzed (Participants) | 891 | 297
  Malaise; Post-Any Injection | 41.8 | 35.4
  Grade 3 Malaise; Post-Any Injection: number analyzed (Participants) | 891 | 297
  Grade 3 Malaise; Post-Any Injection | 4.3 | 2.7
  Myalgia; Post-Any Injection: number analyzed (Participants) | 891 | 297
  Myalgia; Post-Any Injection | 44.2 | 43.8
  Grade 3 Myalgia; Post-Any Injection: number analyzed (Participants) | 891 | 297
  Grade 3 Myalgia; Post-Any Injection | 2.6 | 2.0
  Asthenia; Post-Any Injection: number analyzed (Participants) | 891 | 297
  Asthenia; Post-Any Injection | 20.5 | 17.5
  Grade 3 Asthenia; Post-Any Injection: number analyzed (Participants) | 891 | 297
  Grade 3 Asthenia; Post-Any Injection | 1.3 | 0.7
  Fever; Post-Injection 1: number analyzed (Participants) | 891 | 297
  Fever; Post-Injection 1 | 4.6 | 2.7
  Grade 3 Fever; Post-Injection 1: number analyzed (Participants) | 891 | 297
  Grade 3 Fever; Post-Injection 1 | 0.6 | 0.7
  Headache; Post-Injection 1: number analyzed (Participants) | 891 | 297
  Headache; Post-Injection 1 | 30.0 | 27.3
  Grade 3 Headache; Post-Injection 1: number analyzed (Participants) | 891 | 297
  Grade 3 Headache; Post-Injection 1 | 2.4 | 1.3
  Malaise; Post-Injection 1: number analyzed (Participants) | 891 | 297
  Malaise; Post-Injection 1 | 25.0 | 18.2
  Grade 3 Malaise; Post-Injection 1: number analyzed (Participants) | 891 | 297
  Grade 3 Malaise; Post-Injection 1 | 2.0 | 0.7
  Myalgia; Post-Injection 1: number analyzed (Participants) | 891 | 297
  Myalgia; Post-Injection 1 | 29.4 | 19.2
  Grade 3 Myalgia; Post-Injection 1: number analyzed (Participants) | 891 | 297
  Grade 3 Myalgia; Post-Injection 1 | 1.3 | 1.0
  Asthenia; Post-Injection 1: number analyzed (Participants) | 891 | 297
  Asthenia; Post-Injection 1 | 12.8 | 6.1
  Grade 3 Asthenia; Post-Injection 1: number analyzed (Participants) | 891 | 297
  Grade 3 Asthenia; Post-Injection 1 | 0.7 | 0.3
  Fever; Post-Injection 2: number analyzed (Participants) | 859 | 285
  Fever; Post-Injection 2 | 3.3 | 2.8
  Grade 3 Fever; Post-Injection 2: number analyzed (Participants) | 859 | 285
  Grade 3 Fever; Post-Injection 2 | 0.6 | 0.0
  Headache; Post-Injection 2: number analyzed (Participants) | 859 | 285
  Headache; Post-Injection 2 | 22.8 | 21.8
  Grade 3 Headache; Post-Injection 2: number analyzed (Participants) | 859 | 285
  Grade 3 Headache; Post-Injection 2 | 0.7 | 1.1
  Malaise; Post-Injection 2: number analyzed (Participants) | 859 | 285
  Malaise; Post-Injection 2 | 19.1 | 18.2
  Grade 3 Malaise; Post-Injection 2: number analyzed (Participants) | 859 | 285
  Grade 3 Malaise; Post-Injection 2 | 1.2 | 1.1
  Myalgia; Post-Injection 2: number analyzed (Participants) | 859 | 285
  Myalgia; Post-Injection 2 | 24.0 | 29.5
  Grade 3 Myalgia; Post-Injection 2: number analyzed (Participants) | 859 | 285
  Grade 3 Myalgia; Post-Injection 2 | 0.9 | 0.7
  Asthenia; Post-Injection 2: number analyzed (Participants) | 859 | 285
  Asthenia; Post-Injection 2 | 9.3 | 10.2
  Grade 3 Asthenia; Post-Injection 2: number analyzed (Participants) | 859 | 285
  Grade 3 Asthenia; Post-Injection 2 | 0.3 | 0.0
  Fever; Post-Injection 3: number analyzed (Participants) | 836 | 278
  Fever; Post-Injection 3 | 4.8 | 2.9
  Grade 3 Fever; Post-Injection 3: number analyzed (Participants) | 836 | 278
  Grade 3 Fever; Post-Injection 3 | 0.8 | 0.4
  Headache; Post-Injection 3: number analyzed (Participants) | 836 | 278
  Headache; Post-Injection 3 | 20.1 | 19.8
  Grade 3 Headache; Post-Injection 3: number analyzed (Participants) | 836 | 278
  Grade 3 Headache; Post-Injection 3 | 1.0 | 0.4
  Malaise; Post-Injection 3: number analyzed (Participants) | 836 | 278
  Malaise; Post-Injection 3 | 18.2 | 17.3
  Grade 3 Malaise; Post-Injection 3: number analyzed (Participants) | 836 | 278
  Grade 3 Malaise; Post-Injection 3 | 1.4 | 1.1
  Myalgia; Post-Injection 3: number analyzed (Participants) | 836 | 278
  Myalgia; Post-Injection 3 | 21.8 | 26.3
  Grade 3 Myalgia; Post-Injection 3: number analyzed (Participants) | 836 | 278
  Grade 3 Myalgia; Post-Injection 3 | 0.5 | 0.7
  Asthenia; Post-Injection 3: number analyzed (Participants) | 836 | 278
  Asthenia; Post-Injection 3 | 8.5 | 9.4
  Grade 3 Asthenia; Post-Injection 3: number analyzed (Participants) | 836 | 278
  Grade 3 Asthenia; Post-Injection 3 | 0.4 | 0.4

2. Primary Outcome: Percentage of Participants by Age Group (2-11 Years, 12-17 Years, 18-45 Years) Reporting Solicited Injection-site and Systemic Reactions Following Each Injection (Inj.) With CYD Dengue Vaccine or Placebo
Description: Solicited injection site reactions: Pain, Erythema, and Swelling. Solicited systemic reactions: Fever, Headache, Malaise, Myalgia, and Asthenia.
Time Frame: Day 0 up to 14 days post-each injection
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 898 | 300
Percentage of participants
  2-11 years; Injection site Pain, Post-Inj. 1: number analyzed (Participants) | 236 | 80
  2-11 years; Injection site Pain, Post-Inj. 1 | 33.9 | 30.0
  2-11 years; Inj. site Erythema, Post-Inj. 1: number analyzed (Participants) | 236 | 80
  2-11 years; Inj. site Erythema, Post-Inj. 1 | 6.4 | 7.5
  2-11 years; Inj. site Swelling, Post-Inj. 1: number analyzed (Participants) | 236 | 80
  2-11 years; Inj. site Swelling, Post-Inj. 1 | 3.8 | 6.3
  12-17 years; Injection site Pain, Post- Inj. 1: number analyzed (Participants) | 141 | 46
  12-17 years; Injection site Pain, Post- Inj. 1 | 28.4 | 28.3
  12-17 years; Inj. site Erythema, Post- Inj. 1: number analyzed (Participants) | 140 | 46
  12-17 years; Inj. site Erythema, Post- Inj. 1 | 0.0 | 0.0
  12-17 years; Inj. site Swelling, Post-Inj. 1: number analyzed (Participants) | 141 | 46
  12-17 years; Inj. site Swelling, Post-Inj. 1 | 0.0 | 0.0
  18-45 years; Injection site Pain, Post- Inj. 1: number analyzed (Participants) | 515 | 171
  18-45 years; Injection site Pain, Post- Inj. 1 | 30.9 | 16.4
  18-45 years; Inj. site Erythema, Post- Inj. 1: number analyzed (Participants) | 515 | 171
  18-45 years; Inj. site Erythema, Post- Inj. 1 | 0.6 | 0.0
  18-45 years; Inj. site Swelling, Post-Inj. 1: number analyzed (Participants) | 515 | 171
  18-45 years; Inj. site Swelling, Post-Inj. 1 | 0.2 | 0.0
  2-11 years; Injection site Pain, Post- Inj. 2: number analyzed (Participants) | 235 | 76
  2-11 years; Injection site Pain, Post- Inj. 2 | 38.3 | 42.1
  2-11 years; Inj. site Erythema, Post-Inj. 2: number analyzed (Participants) | 235 | 76
  2-11 years; Inj. site Erythema, Post-Inj. 2 | 9.4 | 5.3
  2-11 years; Inj. site Swelling, Post-Inj. 2: number analyzed (Participants) | 235 | 76
  2-11 years; Inj. site Swelling, Post-Inj. 2 | 4.7 | 3.9
  12-17 years; Injection site Pain, Post- Inj. 2: number analyzed (Participants) | 136 | 45
  12-17 years; Injection site Pain, Post- Inj. 2 | 29.4 | 44.4
  12-17 years; Inj. site Erythema, Post- Inj. 2: number analyzed (Participants) | 136 | 45
  12-17 years; Inj. site Erythema, Post- Inj. 2 | 0.0 | 0.0
  12-17 years; Inj. site Swelling, Post-Inj. 2: number analyzed (Participants) | 136 | 45
  12-17 years; Inj. site Swelling, Post-Inj. 2 | 0.0 | 0.0
  18-45 years; Injection site Pain, Post- Inj. 2: number analyzed (Participants) | 488 | 164
  18-45 years; Injection site Pain, Post- Inj. 2 | 38.3 | 62.8
  18-45 years; Inj. site Erythema, Post- Inj. 2: number analyzed (Participants) | 488 | 164
  18-45 years; Inj. site Erythema, Post- Inj. 2 | 1.4 | 12.8
  18-45 years; Inj. site Swelling, Post-Inj. 2: number analyzed (Participants) | 488 | 164
  18-45 years; Inj. site Swelling, Post-Inj. 2 | 0.2 | 4.3
  2-11 years; Injection site Pain, Post- Inj. 3: number analyzed (Participants) | 233 | 76
  2-11 years; Injection site Pain, Post- Inj. 3 | 32.6 | 34.2
  2-11 years; Inj. site Erythema, Post-Inj. 3: number analyzed (Participants) | 233 | 76
  2-11 years; Inj. site Erythema, Post-Inj. 3 | 8.2 | 6.6
  2-11 years; Inj. site Swelling, Post-Inj. 3: number analyzed (Participants) | 233 | 76
  2-11 years; Inj. site Swelling, Post-Inj. 3 | 6.4 | 2.6
  12-17 years; Injection site Pain, Post- Inj. 3: number analyzed (Participants) | 135 | 44
  12-17 years; Injection site Pain, Post- Inj. 3 | 26.7 | 38.6
  12-17 years; Inj. site Erythema, Post- Inj. 3: number analyzed (Participants) | 135 | 44
  12-17 years; Inj. site Erythema, Post- Inj. 3 | 0.0 | 0.0
  12-17 years; Inj. site Swelling, Post-Inj. 3: number analyzed (Participants) | 135 | 44
  12-17 years; Inj. site Swelling, Post-Inj. 3 | 0.0 | 0.0
  18-45 years; Injection site Pain, Post- Inj. 3: number analyzed (Participants) | 468 | 158
  18-45 years; Injection site Pain, Post- Inj. 3 | 38.5 | 60.8
  18-45 years; Inj. site Erythema, Post- Inj. 3: number analyzed (Participants) | 468 | 158
  18-45 years; Inj. site Erythema, Post- Inj. 3 | 2.8 | 13.3
  18-45 years; Inj. site Swelling, Post-Inj. 3: number analyzed (Participants) | 468 | 158
  18-45 years; Inj. site Swelling, Post-Inj. 3 | 1.5 | 8.9
  2-11 years; Fever, Post-Inj. 1: number analyzed (Participants) | 236 | 80
  2-11 years; Fever, Post-Inj. 1 | 8.1 | 6.3
  2-11 years; Headache, Post-Inj. 1: number analyzed (Participants) | 236 | 80
  2-11 years; Headache, Post-Inj. 1 | 25.0 | 16.3
  2-11 years; Malaise, Post-Inj. 1: number analyzed (Participants) | 236 | 80
  2-11 years; Malaise, Post-Inj. 1 | 19.9 | 13.8
  2-11 years; Myalgia, Post-Inj. 1: number analyzed (Participants) | 236 | 80
  2-11 years; Myalgia, Post-Inj. 1 | 23.7 | 16.3
  2-11 years; Asthenia, Post-Inj. 1: number analyzed (Participants) | 236 | 80
  2-11 years; Asthenia, Post-Inj. 1 | 7.2 | 3.8
  12-17 years; Fever, Post-Inj. 1: number analyzed (Participants) | 140 | 46
  12-17 years; Fever, Post-Inj. 1 | 7.1 | 2.2
  12-17 years; Headache, Post-Inj. 1: number analyzed (Participants) | 140 | 46
  12-17 years; Headache, Post-Inj. 1 | 39.3 | 39.1
  12-17 years; Malaise, Post-Inj. 1: number analyzed (Participants) | 140 | 46
  12-17 years; Malaise, Post-Inj. 1 | 29.3 | 17.4
  12-17 years; Myalgia, Post-Inj. 1: number analyzed (Participants) | 140 | 46
  12-17 years; Myalgia, Post-Inj. 1 | 32.1 | 23.9
  12-17 years; Asthenia, Post-Inj. 1: number analyzed (Participants) | 140 | 46
  12-17 years; Asthenia, Post-Inj. 1 | 13.6 | 6.5
  18-45 years; Fever, Post-Inj. 1: number analyzed (Participants) | 515 | 171
  18-45 years; Fever, Post-Inj. 1 | 2.3 | 1.2
  18-45 years; Headache, Post-Inj. 1: number analyzed (Participants) | 515 | 171
  18-45 years; Headache, Post-Inj. 1 | 29.7 | 29.2
  18-45 years; Malaise, Post-Inj. 1: number analyzed (Participants) | 515 | 171
  18-45 years; Malaise, Post-Inj. 1 | 26.2 | 20.5
  18-45 years; Myalgia, Post-Inj. 1: number analyzed (Participants) | 515 | 171
  18-45 years; Myalgia, Post-Inj. 1 | 31.3 | 19.3
  18-45 years; Asthenia, Post-Inj. 1: number analyzed (Participants) | 515 | 171
  18-45 years; Asthenia, Post-Inj. 1 | 15.1 | 7.0
  2-11 years; Fever, Post-Inj. 2: number analyzed (Participants) | 235 | 76
  2-11 years; Fever, Post-Inj. 2 | 6.8 | 6.6
  2-11 years; Headache, Post-Inj. 2: number analyzed (Participants) | 235 | 76
  2-11 years; Headache, Post-Inj. 2 | 21.7 | 15.8
  2-11 years; Malaise, Post-Inj. 2: number analyzed (Participants) | 235 | 76
  2-11 years; Malaise, Post-Inj. 2 | 21.7 | 13.2
  2-11 years; Myalgia, Post-Inj. 2: number analyzed (Participants) | 235 | 76
  2-11 years; Myalgia, Post-Inj. 2 | 24.7 | 22.4
  2-11 years; Asthenia, Post-Inj. 2: number analyzed (Participants) | 235 | 76
  2-11 years; Asthenia, Post-Inj. 2 | 7.7 | 7.9
  12-17 years; Fever, Post-Inj. 2: number analyzed (Participants) | 136 | 45
  12-17 years; Fever, Post-Inj. 2 | 4.4 | 0.0
  12-17 years; Headache, Post-Inj. 2: number analyzed (Participants) | 136 | 45
  12-17 years; Headache, Post-Inj. 2 | 19.9 | 22.2
  12-17 years; Malaise, Post-Inj. 2: number analyzed (Participants) | 136 | 45
  12-17 years; Malaise, Post-Inj. 2 | 16.2 | 20.0
  12-17 years; Myalgia, Post-Inj. 2: number analyzed (Participants) | 136 | 45
  12-17 years; Myalgia, Post-Inj. 2 | 19.9 | 28.9
  12-17 years; Asthenia, Post-Inj. 2: number analyzed (Participants) | 136 | 45
  12-17 years; Asthenia, Post-Inj. 2 | 8.8 | 6.7
  18-45 years; Fever, Post-Inj. 2: number analyzed (Participants) | 488 | 164
  18-45 years; Fever, Post-Inj. 2 | 1.2 | 1.8
  18-45 years; Headache, Post-Inj. 2: number analyzed (Participants) | 488 | 164
  18-45 years; Headache, Post-Inj. 2 | 24.2 | 24.4
  18-45 years; Malaise, Post-Inj. 2: number analyzed (Participants) | 488 | 164
  18-45 years; Malaise, Post-Inj. 2 | 18.6 | 20.1
  18-45 years; Myalgia, Post-Inj. 2: number analyzed (Participants) | 488 | 164
  18-45 years; Myalgia, Post-Inj. 2 | 24.8 | 32.9
  18-45 years; Asthenia, Post-Inj. 2: number analyzed (Participants) | 488 | 164
  18-45 years; Asthenia, Post-Inj. 2 | 10.2 | 12.2
  2-11 years; Fever, Post-Inj. 3: number analyzed (Participants) | 233 | 76
  2-11 years; Fever, Post-Inj. 3 | 8.2 | 6.6
  2-11 years; Headache, Post-Inj. 3: number analyzed (Participants) | 233 | 76
  2-11 years; Headache, Post-Inj. 3 | 17.6 | 11.8
  2-11 years; Malaise, Post-Inj. 3: number analyzed (Participants) | 233 | 76
  2-11 years; Malaise, Post-Inj. 3 | 18.5 | 14.5
  2-11 years; Myalgia, Post-Inj. 3: number analyzed (Participants) | 233 | 76
  2-11 years; Myalgia, Post-Inj. 3 | 20.6 | 17.1
  2-11 years; Asthenia, Post-Inj. 3: number analyzed (Participants) | 233 | 76
  2-11 years; Asthenia, Post-Inj. 3 | 7.7 | 3.9
  12-17 years; Fever, Post-Inj. 3: number analyzed (Participants) | 135 | 44
  12-17 years; Fever, Post-Inj. 3 | 5.9 | 2.3
  12-17 years; Headache, Post-Inj. 3: number analyzed (Participants) | 135 | 44
  12-17 years; Headache, Post-Inj. 3 | 20.7 | 20.5
  12-17 years; Malaise, Post-Inj. 3: number analyzed (Participants) | 135 | 44
  12-17 years; Malaise, Post-Inj. 3 | 18.5 | 18.2
  12-17 years; Myalgia, Post-Inj. 3: number analyzed (Participants) | 135 | 44
  12-17 years; Myalgia, Post-Inj. 3 | 14.8 | 25.0
  12-17 years; Asthenia, Post-Inj. 3: number analyzed (Participants) | 135 | 44
  12-17 years; Asthenia, Post-Inj. 3 | 5.9 | 11.4
  18-45 years; Fever, Post-Inj. 3: number analyzed (Participants) | 468 | 158
  18-45 years; Fever, Post-Inj. 3 | 2.8 | 1.3
  18-45 years; Headache, Post-Inj. 3: number analyzed (Participants) | 468 | 158
  18-45 years; Headache, Post-Inj. 3 | 21.2 | 23.4
  18-45 years; Malaise, Post-Inj. 3: number analyzed (Participants) | 468 | 158
  18-45 years; Malaise, Post-Inj. 3 | 17.9 | 18.4
  18-45 years; Myalgia, Post-Inj. 3: number analyzed (Participants) | 468 | 158
  18-45 years; Myalgia, Post-Inj. 3 | 24.4 | 31.0
  18-45 years; Asthenia, Post-Inj. 3: number analyzed (Participants) | 468 | 158
  18-45 years; Asthenia, Post-Inj. 3 | 9.6 | 11.4

3. Primary Outcome: Percentage of All Participants Who Achieved Seropositivity Against Each of the Dengue Virus Serotypes Before and After Each Vaccination With CYD Dengue Vaccine or Placebo
Description: Seropositivity against each dengue virus serotype (parental strains) was assessed using a dengue plaque reduction neutralization test (PRNT) assay. Seropositive participants were defined as participants with neutralizing antibody titers >=10 (1/dilution).
Time Frame: Pre-Injection 1, 2, and 3 and 28 days Post-Injection 1, 2, and 3
Population: Analysis was performed on Per-Protocol (PP) analysis set which included all participants who were vaccinated and had no protocol deviations. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 424 | 140
Percentage of participants
  CYD dengue Serotype 1; Pre-Injection 1 | 14.6 | 17.1
  CYD dengue Serotype 1; Post-Injection 1: number analyzed (Participants) | 210 | 69
  CYD dengue Serotype 1; Post-Injection 1 | 22.9 | 11.6
  CYD dengue Serotype 1; Pre-Injection 2: number analyzed (Participants) | 183 | 60
  CYD dengue Serotype 1; Pre-Injection 2 | 30.1 | 16.7
  CYD dengue Serotype 1; Post-Injection 2: number analyzed (Participants) | 184 | 60
  CYD dengue Serotype 1; Post-Injection 2 | 54.9 | 18.3
  CYD dengue Serotype 1; Pre-Injection 3: number analyzed (Participants) | 179 | 58
  CYD dengue Serotype 1; Pre-Injection 3 | 45.8 | 13.8
  CYD dengue Serotype 1; Post-Injection 3: number analyzed (Participants) | 353 | 101
  CYD dengue Serotype 1; Post-Injection 3 | 79.6 | 22.0
  CYD dengue Serotype 2; Pre-Injection 1: number analyzed (Participants) | 422 | 140
  CYD dengue Serotype 2; Pre-Injection 1 | 16.1 | 15.0
  CYD dengue Serotype 2; Post-Injection 1: number analyzed (Participants) | 210 | 69
  CYD dengue Serotype 2; Post-Injection 1 | 39.5 | 10.1
  CYD dengue Serotype 2; Pre-Injection 2: number analyzed (Participants) | 183 | 60
  CYD dengue Serotype 2; Pre-Injection 2 | 39.3 | 16.7
  CYD dengue Serotype 2; Post-Injection 2: number analyzed (Participants) | 184 | 60
  CYD dengue Serotype 2; Post-Injection 2 | 80.4 | 15.0
  CYD dengue Serotype 2; Pre-Injection 3: number analyzed (Participants) | 180 | 58
  CYD dengue Serotype 2; Pre-Injection 3 | 58.3 | 13.8
  CYD dengue Serotype 2; Post-Injection 3: number analyzed (Participants) | 353 | 109
  CYD dengue Serotype 2; Post-Injection 3 | 88.1 | 20.2
  CYD dengue Serotype 3; Pre-Injection 1: number analyzed (Participants) | 421 | 139
  CYD dengue Serotype 3; Pre-Injection 1 | 19.7 | 20.1
  CYD dengue Serotype 3; Post-Injection 1: number analyzed (Participants) | 208 | 69
  CYD dengue Serotype 3; Post-Injection 1 | 58.7 | 21.7
  CYD dengue Serotype 3; Pre-Injection 2: number analyzed (Participants) | 183 | 58
  CYD dengue Serotype 3; Pre-Injection 2 | 63.9 | 31.0
  CYD dengue Serotype 3; Post-Injection 2: number analyzed (Participants) | 183 | 60
  CYD dengue Serotype 3; Post-Injection 2 | 87.4 | 26.7
  CYD dengue Serotype 3; Pre-Injection 3: number analyzed (Participants) | 180 | 58
  CYD dengue Serotype 3; Pre-Injection 3 | 77.8 | 19.0
  CYD dengue Serotype 3; Post-Injection 3: number analyzed (Participants) | 352 | 109
  CYD dengue Serotype 3; Post-Injection 3 | 93.2 | 24.8
  CYD dengue Serotype 4; Pre-Injection 1: number analyzed (Participants) | 421 | 139
  CYD dengue Serotype 4; Pre-Injection 1 | 12.8 | 12.9
  CYD dengue Serotype 4; Post-Injection 1: number analyzed (Participants) | 208 | 69
  CYD dengue Serotype 4; Post-Injection 1 | 67.3 | 11.6
  CYD dengue Serotype 4; Pre-Injection 2: number analyzed (Participants) | 181 | 60
  CYD dengue Serotype 4; Pre-Injection 2 | 69.1 | 16.7
  CYD dengue Serotype 4; Post-Injection 2: number analyzed (Participants) | 183 | 59
  CYD dengue Serotype 4; Post-Injection 2 | 85.8 | 16.9
  CYD dengue Serotype 4; Pre-Injection 3: number analyzed (Participants) | 179 | 58
  CYD dengue Serotype 4; Pre-Injection 3 | 79.3 | 8.6
  CYD dengue Serotype 4; Post-Injection 3: number analyzed (Participants) | 351 | 109
  CYD dengue Serotype 4; Post-Injection 3 | 93.7 | 19.3

4. Primary Outcome: Percentage of Participants by Age Group (2-11 Years, 12-17 Years, 18-45 Years) Who Achieved Seropositivity Against Each of the Dengue Virus Serotypes Before and After the Third Vaccination With CYD Dengue Vaccine or Placebo
Description: Seropositivity against each dengue virus serotypes (parental strains) was assessed using a dengue PRNT assay. Seropositive participants were defined as participants with neutralizing antibody titers >=10 (1/dilution).
Time Frame: Pre-Injection 1 and 28 days Post-Injection 3
Population: Analysis was performed on Per-Protocol analysis set. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure and 'number analyzed' = participants with available data for each specified category.
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 148 | 47
Percentage of participants
  2-11 years, CYD dengue Serotype 1; Pre-Inj. 1 | 4.7 | 8.5
  2-11 years, CYD dengue Serotype 1; Post-Inj. 3: number analyzed (Participants) | 132 | 37
  2-11 years, CYD dengue Serotype 1; Post-Inj. 3 | 92.4 | 10.8
  2-11 years, CYD dengue Serotype 2; Pre-Inj. 1: number analyzed (Participants) | 147 | 47
  2-11 years, CYD dengue Serotype 2; Pre-Inj. 1 | 5.4 | 2.1
  2-11 years, CYD dengue Serotype 2; Post-Inj. 3: number analyzed (Participants) | 132 | 37
  2-11 years, CYD dengue Serotype 2; Post-Inj. 3 | 93.9 | 16.2
  2-11 years, CYD dengue Serotype 3; Pre-Inj. 1: number analyzed (Participants) | 147 | 47
  2-11 years, CYD dengue Serotype 3; Pre-Inj. 1 | 11.6 | 10.6
  2-11 years, CYD dengue Serotype 3; Post-Inj. 3: number analyzed (Participants) | 132 | 37
  2-11 years, CYD dengue Serotype 3; Post-Inj. 3 | 98.5 | 13.5
  2-11 years, CYD dengue Serotype 4; Pre-Inj. 1 | 6.8 | 6.4
  2-11 years, CYD dengue Serotype 4; Post-Inj. 3: number analyzed (Participants) | 131 | 37
  2-11 years, CYD dengue Serotype 4; Post-Inj. 3 | 96.9 | 18.9
  12-17 years, CYD dengue Serotype 1; Pre-Inj. 1: number analyzed (Participants) | 140 | 46
  12-17 years, CYD dengue Serotype 1; Pre-Inj. 1 | 5.7 | 4.3
  12-17 years, CYD dengue Serotype 1; Post-Inj. 3: number analyzed (Participants) | 123 | 38
  12-17 years, CYD dengue Serotype 1; Post-Inj. 3 | 68.3 | 13.2
  12-17 years, CYD dengue Serotype 2; Pre-Inj. 1: number analyzed (Participants) | 140 | 46
  12-17 years, CYD dengue Serotype 2; Pre-Inj. 1 | 10.0 | 4.3
  12-17 years, CYD dengue Serotype 2; Post-Inj. 3: number analyzed (Participants) | 123 | 38
  12-17 years, CYD dengue Serotype 2; Post-Inj. 3 | 87.0 | 10.5
  12-17 years, CYD dengue Serotype 3; Pre-Inj. 1: number analyzed (Participants) | 139 | 46
  12-17 years, CYD dengue Serotype 3; Pre-Inj. 1 | 11.5 | 10.9
  12-17 years, CYD dengue Serotype 3; Post-Inj. 3: number analyzed (Participants) | 122 | 38
  12-17 years, CYD dengue Serotype 3; Post-Inj. 3 | 88.5 | 21.1
  12-17 years, CYD dengue Serotype 4; Pre-Inj. 1: number analyzed (Participants) | 139 | 46
  12-17 years, CYD dengue Serotype 4; Pre-Inj. 1 | 6.5 | 2.2
  12-17 years, CYD dengue Serotype 4; Post-Inj. 3: number analyzed (Participants) | 123 | 38
  12-17 years, CYD dengue Serotype 4; Post-Inj. 3 | 91.1 | 10.5
  18-45 years, CYD dengue Serotype 1; Pre-Inj. 1: number analyzed (Participants) | 136 | 47
  18-45 years, CYD dengue Serotype 1; Pre-Inj. 1 | 34.6 | 38.3
  18-45 years, CYD dengue Serotype 1; Post-Inj. 3: number analyzed (Participants) | 98 | 34
  18-45 years, CYD dengue Serotype 1; Post-Inj. 3 | 76.5 | 44.1
  18-45 years, CYD dengue Serotype 2; Pre-Inj. 1: number analyzed (Participants) | 135 | 47
  18-45 years, CYD dengue Serotype 2; Pre-Inj. 1 | 34.1 | 38.3
  18-45 years, CYD dengue Serotype 2; Post-Inj. 3: number analyzed (Participants) | 98 | 34
  18-45 years, CYD dengue Serotype 2; Post-Inj. 3 | 81.6 | 35.3
  18-45 years, CYD dengue Serotype 3; Pre-Inj. 1: number analyzed (Participants) | 135 | 46
  18-45 years, CYD dengue Serotype 3; Pre-Inj. 1 | 37.0 | 39.1
  18-45 years, CYD dengue Serotype 3; Post-Inj. 3: number analyzed (Participants) | 98 | 34
  18-45 years, CYD dengue Serotype 3; Post-Inj. 3 | 91.8 | 41.2
  18-45 years, CYD dengue Serotype 4; Pre-Inj. 1: number analyzed (Participants) | 134 | 46
  18-45 years, CYD dengue Serotype 4; Pre-Inj. 1 | 26.1 | 30.4
  18-45 years, CYD dengue Serotype 4; Post-Inj. 3: number analyzed (Participants) | 97 | 34
  18-45 years, CYD dengue Serotype 4; Post-Inj. 3 | 92.8 | 29.4

5. Primary Outcome: Percentage of Participants by Age Group (2-11 Years, 12-17 Years, 18-45 Years) Who Achieved Seropositivity Against at Least 1, 2, 3, or 4 of the Dengue Virus Serotypes Before and After the Third Vaccination With CYD Dengue Vaccine or Placebo
Description: Seropositivity against at least 1, 2, 3, or 4 dengue virus serotypes (parental strains) was assessed using a dengue PRNT assay. Seropositive participants were defined as participants with neutralizing antibody titers >=10 (1/dilution).
Time Frame: Pre-Injection 1 and 28 days Post-Injection 3
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 148 | 47
Percentage of participants
  2-11 yrs, CYD dengue >=1 serotype; Pre- Inj. 1 | 19.6 | 27.7
  2-11 yrs, CYD dengue >=1 serotype; Post-Inj. 3: number analyzed (Participants) | 132 | 37
  2-11 yrs, CYD dengue >=1 serotype; Post-Inj. 3 | 100 | 56.8
  2-11 yrs, CYD dengue >=2 serotypes; Pre-Inj. 1 | 6.1 | 0.0
  2-11 yrs, CYD dengue >=2 serotypes; Post-Inj. 3: number analyzed (Participants) | 132 | 37
  2-11 yrs, CYD dengue >=2 serotypes; Post-Inj. 3 | 99.2 | 2.7
  2-11 yrs, CYD dengue >=3 serotypes; Pre-Inj. 1 | 2.0 | 0.0
  2-11 yrs, CYD dengue >=3 serotypes; Post-Inj. 3: number analyzed (Participants) | 132 | 37
  2-11 yrs, CYD dengue >=3 serotypes; Post-Inj. 3 | 97.0 | 0.0
  2-11 yrs, CYD dengue All 4 serotypes; Pre-Inj. 1 | 0.7 | 0.0
  2-11 yrs, CYD dengue All 4 serotypes; Post-Inj. 3: number analyzed (Participants) | 132 | 37
  2-11 yrs, CYD dengue All 4 serotypes; Post-Inj. 3 | 84.8 | 0.0
  12-17 yrs, CYD dengue >=1 serotype; Pre-Inj. 1: number analyzed (Participants) | 140 | 46
  12-17 yrs, CYD dengue >=1 serotype; Pre-Inj. 1 | 13.6 | 15.2
  12-17 yrs, CYD dengue >=1 serotype; Post-Inj. 3: number analyzed (Participants) | 123 | 38
  12-17 yrs, CYD dengue >=1 serotype; Post-Inj. 3 | 98.4 | 26.3
  12-17 yrs, CYD dengue >=2 serotypes; Pre-Inj. 1: number analyzed (Participants) | 140 | 46
  12-17 yrs, CYD dengue >=2 serotypes; Pre-Inj. 1 | 7.9 | 4.3
  12-17 yrs, CYD dengue >=2 serotypes; Post-Inj. 3: number analyzed (Participants) | 123 | 38
  12-17 yrs, CYD dengue >=2 serotypes; Post-Inj. 3 | 95.1 | 10.5
  12-17 yrs, CYD dengue >=3 serotypes; Pre-Inj. 1: number analyzed (Participants) | 140 | 46
  12-17 yrs, CYD dengue >=3 serotypes; Pre-Inj. 1 | 7.1 | 2.2
  12-17 yrs, CYD dengue >=3 serotypes; Post-Inj. 3: number analyzed (Participants) | 123 | 38
  12-17 yrs, CYD dengue >=3 serotypes; Post-Inj. 3 | 81.3 | 10.5
  12-17 yrs, CYD dengue All 4 serotypes; Pre-Inj. 1: number analyzed (Participants) | 140 | 46
  12-17 yrs, CYD dengue All 4 serotypes; Pre-Inj. 1 | 5.0 | 0.0
  12-17 yrs, CYD dengue All 4 serotypes; Post-Inj. 3: number analyzed (Participants) | 123 | 38
  12-17 yrs, CYD dengue All 4 serotypes; Post-Inj. 3 | 59.3 | 7.9
  18-45 yrs, CYD dengue >=1 serotype; Pre-Inj. 1: number analyzed (Participants) | 136 | 47
  18-45 yrs, CYD dengue >=1 serotype; Pre-Inj. 1 | 47.1 | 53.2
  18-45 yrs, CYD dengue >=1 serotype; Post-Inj. 3: number analyzed (Participants) | 98 | 34
  18-45 yrs, CYD dengue >=1 serotype; Post-Inj. 3 | 100 | 55.9
  18-45 yrs, CYD dengue >=2 serotypes; Pre-Inj. 1: number analyzed (Participants) | 136 | 47
  18-45 yrs, CYD dengue >=2 serotypes; Pre-Inj. 1 | 33.8 | 38.3
  18-45 yrs, CYD dengue >=2 serotypes; Post-Inj. 3: number analyzed (Participants) | 98 | 34
  18-45 yrs, CYD dengue >=2 serotypes; Post-Inj. 3 | 96.9 | 35.3
  18-45 yrs, CYD dengue >=3 serotypes; Pre-Inj. 1: number analyzed (Participants) | 136 | 47
  18-45 yrs, CYD dengue >=3 serotypes; Pre-Inj. 1 | 27.9 | 31.9
  18-45 yrs, CYD dengue >=3 serotypes; Post-Inj. 3: number analyzed (Participants) | 98 | 34
  18-45 yrs, CYD dengue >=3 serotypes; Post-Inj. 3 | 83.7 | 32.4
  18-45 yrs, CYD dengue All 4 serotypes; Pre-Inj. 1: number analyzed (Participants) | 136 | 47
  18-45 yrs, CYD dengue All 4 serotypes; Pre-Inj. 1 | 22.1 | 21.3
  18-45 yrs, CYD dengue All 4 serotypes; Post-Inj. 3: number analyzed (Participants) | 98 | 34
  18-45 yrs, CYD dengue All 4 serotypes; Post-Inj. 3 | 61.2 | 26.5

6. Primary Outcome: Geometric Mean Titers (GMTs) of Antibodies in All Participants Against Each Serotype With the Parental Dengue Virus Strain Before and Following Each Vaccination With CYD Dengue Vaccine or Placebo
Description: GMTs against each serotype with the parental dengue virus strains were assessed using a dengue PRNT assay.
Time Frame: Pre-Injection 1, 2, and 3 and 28 days Post-Injection 1, 2, and 3
Population: Analysis was performed on Per-Protocol analysis set. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dilution)
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 424 | 140
Titers (1/dilution)
  CYD dengue Serotype 1; Pre-Injection 1 | 8.20 [7.20 to 9.33] | 8.23 [6.62 to 10.2]
  CYD dengue Serotype 1; Post-Injection 1: number analyzed (Participants) | 210 | 69
  CYD dengue Serotype 1; Post-Injection 1 | 10.0 [8.06 to 12.4] | 7.09 [5.48 to 9.18]
  CYD dengue Serotype 1; Pre-Injection 2: number analyzed (Participants) | 183 | 60
  CYD dengue Serotype 1; Pre-Injection 2 | 12.9 [9.89 to 16.7] | 7.85 [5.79 to 10.6]
  CYD dengue Serotype 1; Post-Injection 2: number analyzed (Participants) | 184 | 60
  CYD dengue Serotype 1; Post-Injection 2 | 22.4 [17.1 to 29.3] | 7.91 [5.85 to 10.7]
  CYD dengue Serotype 1; Pre-Injection 3: number analyzed (Participants) | 179 | 58
  CYD dengue Serotype 1; Pre-Injection 3 | 18.0 [14.0 to 23.2] | 7.40 [5.54 to 9.88]
  CYD dengue Serotype 1; Post-Injection 3: number analyzed (Participants) | 353 | 109
  CYD dengue Serotype 1; Post-Injection 3 | 46.6 [39.0 to 55.6] | 8.93 [7.08 to 11.3]
  CYD dengue Serotype 2; Pre-Injection 1: number analyzed (Participants) | 422 | 140
  CYD dengue Serotype 2; Pre-Injection 1 | 9.06 [7.86 to 10.4] | 8.48 [6.69 to 10.8]
  CYD dengue Serotype 2; Post-Injection 1: number analyzed (Participants) | 210 | 69
  CYD dengue Serotype 2; Post-Injection 1 | 17.2 [13.3 to 22.2] | 7.39 [5.49 to 9.94]
  CYD dengue Serotype 2; Pre-Injection 2: number analyzed (Participants) | 183 | 60
  CYD dengue Serotype 2; Pre-Injection 2 | 19.1 [14.3 to 25.5] | 9.79 [6.45 to 14.9]
  CYD dengue Serotype 2; Post-Injection 2: number analyzed (Participants) | 184 | 60
  CYD dengue Serotype 2; Post-Injection 2 | 50.3 [39.0 to 65.0] | 9.48 [6.22 to 14.4]
  CYD dengue Serotype 2; Pre-Injection 3: number analyzed (Participants) | 180 | 58
  CYD dengue Serotype 2; Pre-Injection 3 | 24.4 [19.2 to 31.1] | 6.98 [5.38 to 9.07]
  CYD dengue Serotype 2; Post-Injection 3: number analyzed (Participants) | 353 | 109
  CYD dengue Serotype 2; Post-Injection 3 | 72.7 [61.6 to 85.8] | 8.88 [6.90 to 11.4]
  CYD dengue Serotype 3; Pre-Injection 1: number analyzed (Participants) | 421 | 139
  CYD dengue Serotype 3; Pre-Injection 1 | 8.45 [7.54 to 9.47] | 8.93 [7.11 to 11.2]
  CYD dengue Serotype 3; Post-Injection 1: number analyzed (Participants) | 208 | 69
  CYD dengue Serotype 3; Post-Injection 1 | 28.2 [22.0 to 36.3] | 9.56 [6.72 to 13.6]
  CYD dengue Serotype 3; Pre-Injection 2: number analyzed (Participants) | 183 | 58
  CYD dengue Serotype 3; Pre-Injection 2 | 29.7 [23.2 to 38.0] | 11.1 [7.60 to 16.3]
  CYD dengue Serotype 3; Post-Injection 2: number analyzed (Participants) | 183 | 60
  CYD dengue Serotype 3; Post-Injection 2 | 70.8 [56.8 to 88.2] | 10.5 [7.36 to 14.9]
  CYD dengue Serotype 3; Pre-Injection 3: number analyzed (Participants) | 180 | 58
  CYD dengue Serotype 3; Pre-Injection 3 | 39.1 [31.2 to 48.9] | 8.23 [5.88 to 11.5]
  CYD dengue Serotype 3; Post-Injection 3: number analyzed (Participants) | 352 | 109
  CYD dengue Serotype 3; Post-Injection 3 | 100 [86.9 to 116] | 9.52 [7.41 to 12.2]
  CYD dengue Serotype 4; Pre-Injection 1: number analyzed (Participants) | 421 | 139
  CYD dengue Serotype 4; Pre-Injection 1 | 6.93 [6.31 to 7.60] | 6.84 [5.86 to 7.99]
  CYD dengue Serotype 4; Post-Injection 1: number analyzed (Participants) | 208 | 69
  CYD dengue Serotype 4; Post-Injection 1 | 65.9 [49.1 to 88.3] | 6.31 [5.30 to 7.50]
  CYD dengue Serotype 4; Pre-Injection 2: number analyzed (Participants) | 181 | 60
  CYD dengue Serotype 4; Pre-Injection 2 | 47.5 [36.5 to 61.8] | 7.91 [5.91 to 10.6]
  CYD dengue Serotype 4; Post-Injection 2: number analyzed (Participants) | 183 | 59
  CYD dengue Serotype 4; Post-Injection 2 | 90.2 [71.7 to 114] | 8.00 [5.89 to 10.9]
  CYD dengue Serotype 4; Pre-Injection 3: number analyzed (Participants) | 179 | 58
  CYD dengue Serotype 4; Pre-Injection 3 | 47.1 [37.9 to 58.5] | 6.04 [5.09 to 7.17]
  CYD dengue Serotype 4; Post-Injection 3: number analyzed (Participants) | 351 | 109
  CYD dengue Serotype 4; Post-Injection 3 | 99.4 [87.4 to 113] | 7.66 [6.35 to 9.24]

7. Primary Outcome: GMTs of Antibodies by Age Groups (2-11 Years, 12-17 Years, 18-45 Years) Against Each Serotype With the Parental Dengue Virus Strain Before and Following the Third Vaccination With CYD Dengue Vaccine
Description: GMTs against each dengue virus serotype (parental strains) were assessed using a dengue PRNT assay.
Time Frame: Pre-Injection 1 and 28 days Post-Injection 3
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dilution)
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 148 | 47
Titers (1/dilution)
  2-11 years, CYD dengue Serotype 1; Pre-Inj. 1 | 5.33 [5.08 to 5.6] | 5.44 [5.01 to 5.92]
  2-11 years, CYD dengue Serotype 1; Post-Inj. 3: number analyzed (Participants) | 132 | 37
  2-11 years, CYD dengue Serotype 1; Post-Inj. 3 | 60.7 [49.5 to 74.3] | 6.32 [4.92 to 8.13]
  2-11 years, CYD dengue Serotype 2; Pre-Inj. 1: number analyzed (Participants) | 147 | 47
  2-11 years, CYD dengue Serotype 2; Pre-Inj. 1 | 5.85 [5.18 to 6.60] | 5.18 [4.82 to 5.57]
  2-11 years, CYD dengue Serotype 2; Post-Inj. 3: number analyzed (Participants) | 132 | 37
  2-11 years, CYD dengue Serotype 2; Post-Inj. 3 | 95.9 [76.7 to 120] | 6.09 [5.18 to 7.16]
  2-11 years, CYD dengue Serotype 3; Pre-Inj. 1: number analyzed (Participants) | 147 | 47
  2-11 years, CYD dengue Serotype 3; Pre-Inj. 1 | 6.24 [5.57 to 6.99] | 6.02 [5.04 to 7.17]
  2-11 years, CYD dengue Serotype 3; Post-Inj. 3: number analyzed (Participants) | 132 | 37
  2-11 years, CYD dengue Serotype 3; Post-Inj. 3 | 138 [115 to 165] | 6.67 [5.11 to 8.71]
  2-11 years, CYD dengue Serotype 4; Pre-Inj. 1 | 5.64 [5.20 to 6.11] | 5.42 [4.92 to 5.97]
  2-11 years, CYD dengue Serotype 4; Post-Inj. 3: number analyzed (Participants) | 131 | 37
  2-11 years, CYD dengue Serotype 4; Post-Inj. 3 | 101 [84.6 to 122] | 6.92 [5.47 to 8.76]
  12-17 years, CYD dengue Serotype 1; Pre-Inj. 1: number analyzed (Participants) | 140 | 46
  12-17 years, CYD dengue Serotype 1; Pre-Inj. 1 | 6.49 [5.31 to 7.92] | 5.47 [4.80 to 6.24]
  12-17 years, CYD dengue Serotype 1; Post-Inj. 3: number analyzed (Participants) | 123 | 38
  12-17 years, CYD dengue Serotype 1; Post-Inj. 3 | 28.9 [21.5 to 38.7] | 6.56 [5.14 to 8.37]
  12-17 years, CYD dengue Serotype 2; Pre-Inj. 1: number analyzed (Participants) | 140 | 46
  12-17 years, CYD dengue Serotype 2; Pre-Inj. 1 | 7.47 [5.96 to 9.37] | 5.54 [4.69 to 6.56]
  12-17 years, CYD dengue Serotype 2; Post-Inj. 3: number analyzed (Participants) | 123 | 38
  12-17 years, CYD dengue Serotype 2; Post-Inj. 3 | 54.0 [41.1 to 70.9] | 6.35 [5.03 to 8.00]
  12-17 years, CYD dengue Serotype 3; Pre-Inj. 1: number analyzed (Participants) | 139 | 46
  12-17 years, CYD dengue Serotype 3; Pre-Inj. 1 | 6.86 [5.82 to 8.09] | 6.83 [4.84 to 9.65]
  12-17 years, CYD dengue Serotype 3; Post-Inj. 3: number analyzed (Participants) | 122 | 38
  12-17 years, CYD dengue Serotype 3; Post-Inj. 3 | 74.1 [57.5 to 95.5] | 8.32 [5.57 to 12.4]
  12-17 years, CYD dengue Serotype 4; Pre-Inj. 1: number analyzed (Participants) | 139 | 46
  12-17 years, CYD dengue Serotype 4; Pre-Inj. 1 | 5.83 [5.18 to 6.57] | 5.08 [4.92 to 5.23]
  12-17 years, CYD dengue Serotype 4; Post-Inj. 3: number analyzed (Participants) | 123 | 38
  12-17 years, CYD dengue Serotype 4; Post-Inj. 3 | 80.4 [64.2 to 101] | 6.68 [4.87 to 9.15]
  18-45 years, CYD dengue Serotype 1; Pre-Inj. 1: number analyzed (Participants) | 136 | 47
  18-45 years, CYD dengue Serotype 1; Pre-Inj. 1 | 16.7 [12.2 to 22.8] | 18.5 [10.4 to 32.9]
  18-45 years, CYD dengue Serotype 1; Post-Inj. 3: number analyzed (Participants) | 98 | 34
  18-45 years, CYD dengue Serotype 1; Post-Inj. 3 | 59.5 [38.7 to 91.6] | 18.3 [10.2 to 33.0]
  18-45 years, CYD dengue Serotype 2; Pre-Inj. 1: number analyzed (Participants) | 135 | 47
  18-45 years, CYD dengue Serotype 2; Pre-Inj. 1 | 17.8 [12.8 to 24.7] | 21.1 [11.3 to 39.2]
  18-45 years, CYD dengue Serotype 2; Post-Inj. 3: number analyzed (Participants) | 98 | 34
  18-45 years, CYD dengue Serotype 2; Post-Inj. 3 | 72.7 [49.4 to 107] | 19.5 [9.69 to 39.1]
  18-45 years, CYD dengue Serotype 3; Pre-Inj. 1: number analyzed (Participants) | 135 | 46
  18-45 years, CYD dengue Serotype 3; Pre-Inj. 1 | 14.6 [11.2 to 19] | 17.5 [10.2 to 30.0]
  18-45 years, CYD dengue Serotype 3; Post-Inj. 3: number analyzed (Participants) | 98 | 34
  18-45 years, CYD dengue Serotype 3; Post-Inj. 3 | 94.9 [69.4 to 130] | 16.3 [9.06 to 29.4]
  18-45 years, CYD dengue Serotype 4; Pre-Inj. 1: number analyzed (Participants) | 134 | 46
  18-45 years, CYD dengue Serotype 4; Pre-Inj. 1 | 10.4 [8.22 to 13.2] | 11.7 [7.65 to 17.9]
  18-45 years, CYD dengue Serotype 4; Post-Inj. 3: number analyzed (Participants) | 97 | 34
  18-45 years, CYD dengue Serotype 4; Post-Inj. 3 | 127 [96 to 167] | 9.96 [6.47 to 15.3]

8. Secondary Outcome: Percentage of Participants Aged 2 to 11 Years Who Achieved Seropositivity Against Each of the Dengue Virus Serotypes Before and up to 4 Years After the Third Vaccination With CYD Dengue Vaccine or Placebo
Description: as for outcome 4
Time Frame: Pre-Injection 1, 28 days Post-Injection 3, at 1 year follow up, 2 year follow up, 3 year follow up and 4 year follow up (assessed post-injection 3 during the follow up duration of 4 years)
Population: Full analysis set included participants who received at least 1 dose of CYD dengue vaccine or Placebo, had at least 1 blood sample drawn and valid post-vaccination serology result. Here, 'overall number of participants analyzed'=participants evaluable for outcome measure and 'number analyzed'=participants with available data for specified category.
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 236 | 80
Percentage of participants
  CYD dengue Serotype 1; Pre-Injection 1: number analyzed (Participants) | 148 | 50
  CYD dengue Serotype 1; Pre-Injection 1 | 4.7 | 8.0
  CYD dengue Serotype 1; Post-Injection 3: number analyzed (Participants) | 144 | 45
  CYD dengue Serotype 1; Post-Injection 3 | 91.0 | 8.9
  CYD dengue Serotype 1; 1st year follow up: number analyzed (Participants) | 141 | 44
  CYD dengue Serotype 1; 1st year follow up | 41.8 | 6.8
  CYD dengue Serotype 1; 2nd year follow up: number analyzed (Participants) | 140 | 43
  CYD dengue Serotype 1; 2nd year follow up | 27.1 | 0.0
  CYD dengue Serotype 1; 3rd year follow up: number analyzed (Participants) | 133 | 43
  CYD dengue Serotype 1; 3rd year follow up | 16.5 | 0.0
  CYD dengue Serotype 1; 4th year follow up: number analyzed (Participants) | 136 | 42
  CYD dengue Serotype 1; 4th year follow up | 9.6 | 0.0
  CYD dengue Serotype 2; Pre-Injection 1: number analyzed (Participants) | 147 | 50
  CYD dengue Serotype 2; Pre-Injection 1 | 5.4 | 2.0
  CYD dengue Serotype 2; Post-Injection 3: number analyzed (Participants) | 144 | 45
  CYD dengue Serotype 2; Post-Injection 3 | 94.4 | 13.3
  CYD dengue Serotype 2; 1st year follow up: number analyzed (Participants) | 141 | 45
  CYD dengue Serotype 2; 1st year follow up | 59.6 | 8.9
  CYD dengue Serotype 2; 2nd year follow up: number analyzed (Participants) | 140 | 43
  CYD dengue Serotype 2; 2nd year follow up | 52.1 | 11.6
  CYD dengue Serotype 2; 3rd year follow up: number analyzed (Participants) | 134 | 43
  CYD dengue Serotype 2; 3rd year follow up | 34.3 | 7.0
  CYD dengue Serotype 2; 4th year follow up: number analyzed (Participants) | 130 | 42
  CYD dengue Serotype 2; 4th year follow up | 36.9 | 2.4
  CYD dengue Serotype 3; Pre-Injection 1: number analyzed (Participants) | 147 | 50
  CYD dengue Serotype 3; Pre-Injection 1 | 11.6 | 10.0
  CYD dengue Serotype 3; Post-Injection 3: number analyzed (Participants) | 144 | 44
  CYD dengue Serotype 3; Post-Injection 3 | 97.9 | 13.6
  CYD dengue Serotype 3; 1st year follow up: number analyzed (Participants) | 141 | 44
  CYD dengue Serotype 3; 1st year follow up | 66.0 | 9.1
  CYD dengue Serotype 3; 2nd year follow up: number analyzed (Participants) | 133 | 41
  CYD dengue Serotype 3; 2nd year follow up | 74.4 | 29.3
  CYD dengue Serotype 3; 3rd year follow up: number analyzed (Participants) | 134 | 43
  CYD dengue Serotype 3; 3rd year follow up | 50.0 | 4.7
  CYD dengue Serotype 3; 4th year follow up: number analyzed (Participants) | 130 | 42
  CYD dengue Serotype 3; 4th year follow up | 37.7 | 2.4
  CYD dengue Serotype 4; Pre-Injection 1: number analyzed (Participants) | 148 | 50
  CYD dengue Serotype 4; Pre-Injection 1 | 6.8 | 6.0
  CYD dengue Serotype 4; Post-Injection 3: number analyzed (Participants) | 143 | 44
  CYD dengue Serotype 4; Post-Injection 3 | 97.2 | 20.5
  CYD dengue Serotype 4; 1st year follow up: number analyzed (Participants) | 141 | 43
  CYD dengue Serotype 4; 1st year follow up | 75.2 | 4.7
  CYD dengue Serotype 4; 2nd year follow up: number analyzed (Participants) | 140 | 43
  CYD dengue Serotype 4; 2nd year follow up | 72.9 | 4.7
  CYD dengue Serotype 4; 3rd year follow up: number analyzed (Participants) | 132 | 43
  CYD dengue Serotype 4; 3rd year follow up | 60.6 | 7.0
  CYD dengue Serotype 4; 4th year follow up: number analyzed (Participants) | 136 | 42
  CYD dengue Serotype 4; 4th year follow up | 49.3 | 0.0

9. Secondary Outcome: Percentage of Participants Aged 12 to 17 Years Old Who Achieved Seropositivity Against Each of the Dengue Virus Serotypes Before and up to 4 Years After the Third Vaccination With CYD Dengue Vaccine or Placebo
Description: Seropositivity against each dengue virus serotypes (parental stains) was assessed using a dengue PRNT assay. Seropositive participants were defined as participants with antibody titers >=10 (1/dilution).
Time Frame: as for outcome 8
Population: Analysis was performed on Full analysis set. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure and 'number analyzed' = participants with available data for each specified category.
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 141 | 46
Percentage of participants
  CYD dengue Serotype 1; Pre-Injection 1 | 5.7 | 4.3
  CYD dengue Serotype 1; Post-Injection 3: number analyzed (Participants) | 135 | 43
  CYD dengue Serotype 1; Post-Injection 3 | 67.4 | 11.6
  CYD dengue Serotype 1; 1st year follow up: number analyzed (Participants) | 132 | 41
  CYD dengue Serotype 1; 1st year follow up | 25.8 | 7.3
  CYD dengue Serotype 1; 2nd year follow up: number analyzed (Participants) | 128 | 40
  CYD dengue Serotype 1; 2nd year follow up | 19.5 | 7.5
  CYD dengue Serotype 1; 3rd year follow up: number analyzed (Participants) | 124 | 40
  CYD dengue Serotype 1; 3rd year follow up | 16.1 | 5.0
  CYD dengue Serotype 1; 4th year follow up: number analyzed (Participants) | 118 | 37
  CYD dengue Serotype 1; 4th year follow up | 11.9 | 5.4
  CYD dengue Serotype 2; Pre-Injection 1 | 9.9 | 4.3
  CYD dengue Serotype 2; Post-Injection 3: number analyzed (Participants) | 135 | 43
  CYD dengue Serotype 2; Post-Injection 3 | 83.7 | 9.3
  CYD dengue Serotype 2; 1st year follow up: number analyzed (Participants) | 131 | 41
  CYD dengue Serotype 2; 1st year follow up | 44.3 | 4.9
  CYD dengue Serotype 2; 2nd year follow up: number analyzed (Participants) | 128 | 40
  CYD dengue Serotype 2; 2nd year follow up | 52.3 | 10.0
  CYD dengue Serotype 2; 3rd year follow up: number analyzed (Participants) | 124 | 40
  CYD dengue Serotype 2; 3rd year follow up | 35.5 | 5.0
  CYD dengue Serotype 2; 4th year follow up: number analyzed (Participants) | 116 | 37
  CYD dengue Serotype 2; 4th year follow up | 36.2 | 5.4
  CYD dengue Serotype 3; Pre-Injection 1: number analyzed (Participants) | 140 | 46
  CYD dengue Serotype 3; Pre-Injection 1 | 11.4 | 10.9
  CYD dengue Serotype 3; Post-Injection 3: number analyzed (Participants) | 134 | 43
  CYD dengue Serotype 3; Post-Injection 3 | 88.8 | 20.9
  CYD dengue Serotype 3; 1st year follow up: number analyzed (Participants) | 133 | 40
  CYD dengue Serotype 3; 1st year follow up | 61.7 | 5.0
  CYD dengue Serotype 3; 2nd year follow up: number analyzed (Participants) | 126 | 40
  CYD dengue Serotype 3; 2nd year follow up | 56.3 | 12.5
  CYD dengue Serotype 3; 3rd year follow up: number analyzed (Participants) | 123 | 40
  CYD dengue Serotype 3; 3rd year follow up | 48.8 | 5.0
  CYD dengue Serotype 3; 4th year follow up: number analyzed (Participants) | 118 | 37
  CYD dengue Serotype 3; 4th year follow up | 47.5 | 5.4
  CYD dengue Serotype 4; Pre-Injection 1: number analyzed (Participants) | 140 | 46
  CYD dengue Serotype 4; Pre-Injection 1 | 6.4 | 2.2
  CYD dengue Serotype 4; Post-Injection 3: number analyzed (Participants) | 135 | 43
  CYD dengue Serotype 4; Post-Injection 3 | 91.1 | 9.3
  CYD dengue Serotype 4; 1st year follow up: number analyzed (Participants) | 132 | 41
  CYD dengue Serotype 4; 1st year follow up | 73.5 | 2.4
  CYD dengue Serotype 4; 2nd year follow up: number analyzed (Participants) | 128 | 40
  CYD dengue Serotype 4; 2nd year follow up | 71.1 | 10.0
  CYD dengue Serotype 4; 3rd year follow up: number analyzed (Participants) | 123 | 40
  CYD dengue Serotype 4; 3rd year follow up | 66.7 | 5.0
  CYD dengue Serotype 4; 4th year follow up: number analyzed (Participants) | 118 | 37
  CYD dengue Serotype 4; 4th year follow up | 61.0 | 8.1

10. Secondary Outcome: Percentage of Participants Aged 18 to 45 Years Who Achieved Seropositivity Against Each of the Dengue Virus Serotypes Before and up to 4 Years After the Third Vaccination With CYD Dengue Vaccine or Placebo
Description: Seropositivity against each dengue virus serotypes (parental stains) was assessed using a dengue PRNT assay. Seropositive participants were defined as participants with neutralizing antibody titers >=10 (1/dilution).
Time Frame: as for outcome 8
Population: as for outcome 9
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 521 | 174
Percentage of participants
  CYD dengue Serotype 1; Pre-Injection 1: number analyzed (Participants) | 142 | 49
  CYD dengue Serotype 1; Pre-Injection 1 | 33.1 | 38.8
  CYD dengue Serotype 1; Post-Injection 3: number analyzed (Participants) | 127 | 43
  CYD dengue Serotype 1; Post-Injection 3 | 71.7 | 39.5
  CYD dengue Serotype 1; 1st year follow up: number analyzed (Participants) | 122 | 44
  CYD dengue Serotype 1; 1st year follow up | 45.9 | 31.8
  CYD dengue Serotype 1; 2nd year follow up: number analyzed (Participants) | 117 | 41
  CYD dengue Serotype 1; 2nd year follow up | 43.6 | 34.1
  CYD dengue Serotype 1; 3rd year follow up: number analyzed (Participants) | 114 | 39
  CYD dengue Serotype 1; 3rd year follow up | 40.4 | 30.8
  CYD dengue Serotype 1; 4th year follow up: number analyzed (Participants) | 106 | 38
  CYD dengue Serotype 1; 4th year follow up | 39.6 | 31.6
  CYD dengue Serotype 2; Pre-Injection 1: number analyzed (Participants) | 141 | 49
  CYD dengue Serotype 2; Pre-Injection 1 | 32.6 | 38.8
  CYD dengue Serotype 2; Post-Injection 3: number analyzed (Participants) | 127 | 43
  CYD dengue Serotype 2; Post-Injection 3 | 80.3 | 30.2
  CYD dengue Serotype 2; 1st year follow up: number analyzed (Participants) | 122 | 44
  CYD dengue Serotype 2; 1st year follow up | 66.4 | 40.9
  CYD dengue Serotype 2; 2nd year follow up: number analyzed (Participants) | 117 | 41
  CYD dengue Serotype 2; 2nd year follow up | 68.4 | 34.1
  CYD dengue Serotype 2; 3rd year follow up: number analyzed (Participants) | 114 | 39
  CYD dengue Serotype 2; 3rd year follow up | 55.3 | 35.9
  CYD dengue Serotype 2; 4th year follow up: number analyzed (Participants) | 105 | 38
  CYD dengue Serotype 2; 4th year follow up | 55.2 | 31.6
  CYD dengue Serotype 3; Pre-Injection 1: number analyzed (Participants) | 141 | 48
  CYD dengue Serotype 3; Pre-Injection 1 | 36.9 | 41.7
  CYD dengue Serotype 3; Post-Injection 3: number analyzed (Participants) | 127 | 43
  CYD dengue Serotype 3; Post-Injection 3 | 92.9 | 34.9
  CYD dengue Serotype 3; 1st year follow up: number analyzed (Participants) | 121 | 44
  CYD dengue Serotype 3; 1st year follow up | 68.6 | 38.6
  CYD dengue Serotype 3; 2nd year follow up: number analyzed (Participants) | 117 | 41
  CYD dengue Serotype 3; 2nd year follow up | 77.8 | 46.3
  CYD dengue Serotype 3; 3rd year follow up: number analyzed (Participants) | 112 | 39
  CYD dengue Serotype 3; 3rd year follow up | 67.9 | 35.9
  CYD dengue Serotype 3; 4th year follow up: number analyzed (Participants) | 106 | 37
  CYD dengue Serotype 3; 4th year follow up | 56.6 | 29.7
  CYD dengue Serotype 4; Pre-Injection 1: number analyzed (Participants) | 140 | 48
  CYD dengue Serotype 4; Pre-Injection 1 | 25.0 | 31.3
  CYD dengue Serotype 4; Post-Injection 3: number analyzed (Participants) | 126 | 43
  CYD dengue Serotype 4; Post-Injection 3 | 93.7 | 32.6
  CYD dengue Serotype 4; 1st year follow up: number analyzed (Participants) | 122 | 44
  CYD dengue Serotype 4; 1st year follow up | 86.9 | 29.5
  CYD dengue Serotype 4; 2nd year follow up: number analyzed (Participants) | 117 | 41
  CYD dengue Serotype 4; 2nd year follow up | 81.2 | 24.4
  CYD dengue Serotype 4; 3rd year follow up: number analyzed (Participants) | 114 | 39
  CYD dengue Serotype 4; 3rd year follow up | 79.8 | 20.5
  CYD dengue Serotype 4; 4th year follow up: number analyzed (Participants) | 107 | 38
  CYD dengue Serotype 4; 4th year follow up | 77.6 | 21.1

11. Secondary Outcome: Percentage of Participants Aged 2 to 11 Years Old Who Achieved Seropositivity Against At Least 1, 2, 3, or 4 of the Dengue Virus Serotypes Before and After the Third Vaccination With CYD Dengue Vaccine or Placebo
Description: Seropositivity against at least 1, 2, 3, or 4 dengue virus serotypes was assessed using a dengue PRNT assay. Seropositive participants were defined as participants with neutralizing antibody titers >=10 (1/dilution).
Time Frame: as for outcome 8
Population: as for outcome 9
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 236 | 80
Percentage of participants
  CYD dengue >=1 serotype; Pre-Injection 1: number analyzed (Participants) | 148 | 50
  CYD dengue >=1 serotype; Pre-Injection 1 | 19.6 | 26.0
  CYD dengue >=1 serotype; Post-Injection 3: number analyzed (Participants) | 144 | 45
  CYD dengue >=1 serotype; Post-Injection 3 | 100.0 | 51.1
  CYD dengue >=1 serotype; 1st year follow up: number analyzed (Participants) | 142 | 45
  CYD dengue >=1 serotype; 1st year follow up | 92.3 | 20.0
  CYD dengue >=1 serotype; 2nd year follow up: number analyzed (Participants) | 140 | 43
  CYD dengue >=1 serotype; 2nd year follow up | 95.0 | 34.9
  CYD dengue >=1 serotype; 3rd year follow up: number analyzed (Participants) | 134 | 43
  CYD dengue >=1 serotype; 3rd year follow up | 76.9 | 7.0
  CYD dengue >=1 serotype; 4th year follow up: number analyzed (Participants) | 136 | 42
  CYD dengue >=1 serotype; 4th year follow up | 72.1 | 4.8
  CYD dengue >=2 serotypes; Pre-Injection 1: number analyzed (Participants) | 148 | 50
  CYD dengue >=2 serotypes; Pre-Injection 1 | 6.1 | 0.0
  CYD dengue >=2 serotypes; Post- Injection 3: number analyzed (Participants) | 144 | 45
  CYD dengue >=2 serotypes; Post- Injection 3 | 99.3 | 4.4
  CYD dengue >=2 serotypes; 1st year follow up: number analyzed (Participants) | 142 | 45
  CYD dengue >=2 serotypes; 1st year follow up | 66.2 | 6.7
  CYD dengue >=2 serotypes; 2nd year follow up: number analyzed (Participants) | 140 | 43
  CYD dengue >=2 serotypes; 2nd year follow up | 70.7 | 9.3
  CYD dengue >=2 serotypes; 3rd year follow up: number analyzed (Participants) | 134 | 43
  CYD dengue >=2 serotypes; 3rd year follow up | 48.5 | 7.0
  CYD dengue >=2 serotypes; 4th year follow up: number analyzed (Participants) | 136 | 42
  CYD dengue >=2 serotypes; 4th year follow up | 35.3 | 0.0
  CYD dengue >=3 serotypes; Pre-Injection 1: number analyzed (Participants) | 148 | 50
  CYD dengue >=3 serotypes; Pre-Injection 1 | 2.0 | 0.0
  CYD dengue >=3 serotypes; Post- Injection 3: number analyzed (Participants) | 144 | 45
  CYD dengue >=3 serotypes; Post- Injection 3 | 96.5 | 0.0
  CYD dengue >=3 serotypes; 1st year follow up: number analyzed (Participants) | 142 | 45
  CYD dengue >=3 serotypes; 1st year follow up | 52.8 | 2.2
  CYD dengue >=3 serotypes; 2nd year follow up: number analyzed (Participants) | 140 | 43
  CYD dengue >=3 serotypes; 2nd year follow up | 42.1 | 0.0
  CYD dengue >=3 serotypes; 3rd year follow up: number analyzed (Participants) | 134 | 43
  CYD dengue >=3 serotypes; 3rd year follow up | 23.9 | 4.7
  CYD dengue >=3 serotypes; 4th year follow up: number analyzed (Participants) | 136 | 42
  CYD dengue >=3 serotypes; 4th year follow up | 16.2 | 0.0
  CYD dengue All 4 serotypes; Pre- Injection 1: number analyzed (Participants) | 148 | 50
  CYD dengue All 4 serotypes; Pre- Injection 1 | 0.7 | 0.0
  CYD dengue All 4 serotypes; Post- Injection 3: number analyzed (Participants) | 144 | 45
  CYD dengue All 4 serotypes; Post- Injection 3 | 84.0 | 0.0
  CYD dengue All 4 serotypes; 1st year follow up: number analyzed (Participants) | 142 | 45
  CYD dengue All 4 serotypes; 1st year follow up | 29.6 | 0.0
  CYD dengue All 4 serotypes; 2nd year follow up: number analyzed (Participants) | 140 | 43
  CYD dengue All 4 serotypes; 2nd year follow up | 15.0 | 0.0
  CYD dengue All 4 serotypes; 3rd year follow up: number analyzed (Participants) | 134 | 43
  CYD dengue All 4 serotypes; 3rd year follow up | 11.2 | 0.0
  CYD dengue All 4 serotypes; 4th year follow up: number analyzed (Participants) | 136 | 42
  CYD dengue All 4 serotypes; 4th year follow up | 6.6 | 0.0

12. Secondary Outcome: Percentage of Participants Aged 12 to 17 Years Old Who Achieved Seropositivity Against at Least 1, 2, 3, or 4 of the Dengue Virus Serotypes Before and After the Third Vaccination With CYD Dengue Vaccine or Placebo
Description: as for outcome 11
Time Frame: as for outcome 8
Population: as for outcome 9
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 141 | 46
Percentage of participants
  CYD dengue >=1 Serotype; Pre-Injection 1 | 13.5 | 15.2
  CYD dengue >=1 Serotype; Post- Injection 3: number analyzed (Participants) | 135 | 43
  CYD dengue >=1 Serotype; Post- Injection 3 | 97.8 | 25.6
  CYD dengue >=1 Serotype; 1st year follow up: number analyzed (Participants) | 133 | 41
  CYD dengue >=1 Serotype; 1st year follow up | 94.7 | 7.3
  CYD dengue >=1 Serotype; 2nd year follow up: number analyzed (Participants) | 128 | 40
  CYD dengue >=1 Serotype; 2nd year follow up | 93.0 | 15.0
  CYD dengue >=1 Serotype; 3rd year follow up: number analyzed (Participants) | 124 | 40
  CYD dengue >=1 Serotype; 3rd year follow up | 89.5 | 5.0
  CYD dengue >=1 serotype; 4th year follow up: number analyzed (Participants) | 118 | 37
  CYD dengue >=1 serotype; 4th year follow up | 81.4 | 8.1
  CYD dengue >=2 Serotypes; Pre- Injection 1 | 7.8 | 4.3
  CYD dengue >=2 Serotypes; Post- Injection 3: number analyzed (Participants) | 135 | 43
  CYD dengue >=2 Serotypes; Post- Injection 3 | 94.8 | 9.3
  CYD dengue >=2 Serotypes; 1st year follow up: number analyzed (Participants) | 133 | 41
  CYD dengue >=2 Serotypes; 1st year follow up | 60.2 | 4.9
  CYD dengue >=2 Serotypes; 2nd year follow up: number analyzed (Participants) | 128 | 40
  CYD dengue >=2 Serotypes; 2nd year follow up | 62.5 | 10.0
  CYD dengue >=2 Serotypes; 3rd year follow up: number analyzed (Participants) | 124 | 40
  CYD dengue >=2 Serotypes; 3rd year follow up | 45.2 | 5.0
  CYD dengue >=2 serotypes; 4th year follow up: number analyzed (Participants) | 118 | 37
  CYD dengue >=2 serotypes; 4th year follow up | 44.9 | 5.4
  CYD dengue >=3 Serotypes; Pre- Injection 1 | 7.1 | 2.2
  CYD dengue >=3 Serotypes; Post- Injection 3: number analyzed (Participants) | 135 | 43
  CYD dengue >=3 Serotypes; Post- Injection 3 | 80.7 | 9.3
  CYD dengue >=3 Serotypes; 1st year follow up: number analyzed (Participants) | 133 | 41
  CYD dengue >=3 Serotypes; 1st year follow up | 33.1 | 4.9
  CYD dengue >=3 Serotypes; 2nd year follow up: number analyzed (Participants) | 128 | 40
  CYD dengue >=3 Serotypes; 2nd year follow up | 31.3 | 7.5
  CYD dengue >=3 Serotypes; 3rd year follow up: number analyzed (Participants) | 124 | 40
  CYD dengue >=3 Serotypes; 3rd year follow up | 22.6 | 5.0
  CYD dengue >=3 serotypes; 4th year follow up: number analyzed (Participants) | 118 | 37
  CYD dengue >=3 serotypes; 4th year follow up | 20.3 | 5.4
  CYD dengue All 4 Serotypes; Pre- Injection 1 | 5.0 | 0.0
  CYD dengue All 4 Serotypes; Post- Injection 3: number analyzed (Participants) | 135 | 43
  CYD dengue All 4 Serotypes; Post- Injection 3 | 57.0 | 7.0
  CYD dengue All 4 Serotypes; 1st year follow up: number analyzed (Participants) | 133 | 41
  CYD dengue All 4 Serotypes; 1st year follow up | 15.8 | 2.4
  CYD dengue All 4 Serotypes; 2nd year follow up: number analyzed (Participants) | 128 | 40
  CYD dengue All 4 Serotypes; 2nd year follow up | 11.7 | 7.5
  CYD dengue All 4 Serotypes; 3rd year follow up: number analyzed (Participants) | 124 | 40
  CYD dengue All 4 Serotypes; 3rd year follow up | 8.9 | 5.0
  CYD dengue All 4 serotypes; 4th year follow up: number analyzed (Participants) | 118 | 37
  CYD dengue All 4 serotypes; 4th year follow up | 9.3 | 5.4

13. Secondary Outcome: Percentage of Participants Aged 18 to 45 Years Old Who Achieved Seropositivity Against at Least 1, 2, 3, or 4 of the Dengue Virus Serotypes Before and After the Third Vaccination With CYD Dengue Vaccine or Placebo
Description: as for outcome 11
Time Frame: as for outcome 8
Population: as for outcome 9
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 521 | 174
Percentage of participants
  CYD dengue >=1 Serotype; Pre-Injection 1: number analyzed (Participants) | 142 | 49
  CYD dengue >=1 Serotype; Pre-Injection 1 | 46.5 | 55.1
  CYD dengue >=1 Serotype; Post- Injection 3: number analyzed (Participants) | 127 | 43
  CYD dengue >=1 Serotype; Post- Injection 3 | 100.0 | 53.5
  CYD dengue >=1 Serotype; 1st year follow up: number analyzed (Participants) | 122 | 44
  CYD dengue >=1 Serotype; 1st year follow up | 96.7 | 50.0
  CYD dengue >=1 Serotype; 2nd year follow up: number analyzed (Participants) | 117 | 41
  CYD dengue >=1 Serotype; 2nd year follow up | 96.6 | 56.1
  CYD dengue >=1 Serotype; 3rd year follow up: number analyzed (Participants) | 114 | 39
  CYD dengue >=1 Serotype; 3rd year follow up | 93.0 | 41.0
  CYD dengue >=1 serotype; 4th year follow up: number analyzed (Participants) | 107 | 38
  CYD dengue >=1 serotype; 4th year follow up | 92.5 | 36.8
  CYD dengue >=2 Serotypes; Pre- Injection 1: number analyzed (Participants) | 142 | 49
  CYD dengue >=2 Serotypes; Pre- Injection 1 | 32.4 | 38.8
  CYD dengue >=2 Serotypes; Post- Injection 3: number analyzed (Participants) | 127 | 43
  CYD dengue >=2 Serotypes; Post- Injection 3 | 97.6 | 32.6
  CYD dengue >=2 Serotypes; 1st year follow up: number analyzed (Participants) | 122 | 44
  CYD dengue >=2 Serotypes; 1st year follow up | 73.8 | 38.6
  CYD dengue >=2 Serotypes; 2nd year follow up: number analyzed (Participants) | 117 | 41
  CYD dengue >=2 Serotypes; 2nd year follow up | 76.9 | 34.1
  CYD dengue >=2 Serotypes; 3rd year follow up: number analyzed (Participants) | 114 | 39
  CYD dengue >=2 Serotypes; 3rd year follow up | 63.2 | 33.3
  CYD dengue >=2 serotypes; 4th year follow up: number analyzed (Participants) | 107 | 38
  CYD dengue >=2 serotypes; 4th year follow up | 54.2 | 28.9
  CYD dengue >=3 Serotypes; Pre- Injection 1: number analyzed (Participants) | 142 | 49
  CYD dengue >=3 Serotypes; Pre- Injection 1 | 26.8 | 32.7
  CYD dengue >=3 Serotypes; Post- Injection 3: number analyzed (Participants) | 127 | 43
  CYD dengue >=3 Serotypes; Post- Injection 3 | 83.5 | 27.9
  CYD dengue >=3 Serotypes; 1st year follow up: number analyzed (Participants) | 122 | 44
  CYD dengue >=3 Serotypes; 1st year follow up | 55.7 | 34.1
  CYD dengue >=3 Serotypes; 2nd year follow up: number analyzed (Participants) | 117 | 41
  CYD dengue >=3 Serotypes; 2nd year follow up | 56.4 | 29.3
  CYD dengue >=3 Serotypes; 3rd year follow up: number analyzed (Participants) | 114 | 39
  CYD dengue >=3 Serotypes; 3rd year follow up | 46.5 | 30.8
  CYD dengue >=3 serotypes; 4th year follow up: number analyzed (Participants) | 107 | 38
  CYD dengue >=3 serotypes; 4th year follow up | 43.0 | 26.3
  CYD dengue All 4 Serotypes; Pre- Injection 1: number analyzed (Participants) | 142 | 49
  CYD dengue All 4 Serotypes; Pre- Injection 1 | 21.1 | 22.4
  CYD dengue All 4 Serotypes; Post- Injection 3: number analyzed (Participants) | 127 | 43
  CYD dengue All 4 Serotypes; Post- Injection 3 | 56.7 | 23.3
  CYD dengue All 4 Serotypes; 1st year follow up: number analyzed (Participants) | 122 | 44
  CYD dengue All 4 Serotypes; 1st year follow up | 41.0 | 18.2
  CYD dengue All 4 Serotypes; 2nd year follow up: number analyzed (Participants) | 117 | 41
  CYD dengue All 4 Serotypes; 2nd year follow up | 41.0 | 19.5
  CYD dengue All 4 Serotypes; 3rd year follow up: number analyzed (Participants) | 114 | 39
  CYD dengue All 4 Serotypes; 3rd year follow up | 39.5 | 17.9
  CYD dengue All 4 serotypes; 4th year follow up: number analyzed (Participants) | 107 | 38
  CYD dengue All 4 serotypes; 4th year follow up | 37.4 | 21.1

14. Secondary Outcome: GMTs of Antibodies in Participants 2 to 11 Years Old Against Each Serotype With the Parental Dengue Virus Strain Before and Following the Third Vaccination With CYD Dengue Vaccine
Description: GMTs against each serotype with the dengue virus strain (parental strains) were assessed using a dengue PRNT assay.
Time Frame: as for outcome 8
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dilution)
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 236 | 80
Titers (1/dilution)
  CYD dengue Serotype 1; Pre-Injection 1: number analyzed (Participants) | 148 | 50
  CYD dengue Serotype 1; Pre-Injection 1 | 5.33 [5.08 to 5.60] | 5.42 [5 to 5.86]
  CYD dengue Serotype 1; Post-Injection 3: number analyzed (Participants) | 144 | 45
  CYD dengue Serotype 1; Post-Injection 3 | 56.6 [46.5 to 68.9] | 6.06 [4.93 to 7.46]
  CYD dengue Serotype 1; 1st year follow up: number analyzed (Participants) | 141 | 44
  CYD dengue Serotype 1; 1st year follow up | 12.1 [9.92 to 14.7] | 5.52 [4.92 to 6.19]
  CYD dengue Serotype 1; 2nd year follow up: number analyzed (Participants) | 140 | 43
  CYD dengue Serotype 1; 2nd year follow up | 8.89 [7.5 to 10.5] | 5.00 [5.00 to 5.00]
  CYD dengue Serotype 1; 3rd year follow up: number analyzed (Participants) | 133 | 43
  CYD dengue Serotype 1; 3rd year follow up | 7.35 [6.22 to 8.67] | 5.00 [5.00 to 5.00]
  CYD dengue Serotype 1; 4th year follow up: number analyzed (Participants) | 136 | 42
  CYD dengue Serotype 1; 4th year follow up | 6.21 [5.51 to 7.00] | 5.00 [5.00 to 5.00]
  CYD dengue Serotype 2; Pre-Injection 1: number analyzed (Participants) | 147 | 50
  CYD dengue Serotype 2; Pre-Injection 1 | 5.85 [5.18 to 6.60] | 5.17 [4.83 to 5.53]
  CYD dengue Serotype 2; Post-Injection 3: number analyzed (Participants) | 144 | 45
  CYD dengue Serotype 2; Post-Injection 3 | 101 [81.7 to 125] | 5.88 [5.15 to 6.72]
  CYD dengue Serotype 2; 1st year follow up: number analyzed (Participants) | 141 | 45
  CYD dengue Serotype 2; 1st year follow up | 21.1 [16.6 to 26.9] | 5.86 [4.79 to 7.16]
  CYD dengue Serotype 2; 2nd year follow up: number analyzed (Participants) | 140 | 43
  CYD dengue Serotype 2; 2nd year follow up | 16.4 [12.9 to 20.9] | 6.11 [5.10 to 7.32]
  CYD dengue Serotype 2; 3rd year follow up: number analyzed (Participants) | 134 | 43
  CYD dengue Serotype 2; 3rd year follow up | 11.7 [9.10 to 15.1] | 5.58 [4.86 to 6.41]
  CYD dengue Serotype 2; 4th year follow up: number analyzed (Participants) | 130 | 42
  CYD dengue Serotype 2; 4th year follow up | 14.2 [10.7 to 19.0] | 5.11 [4.89 to 5.32]
  CYD dengue Serotype 3; Pre-Injection 1: number analyzed (Participants) | 147 | 50
  CYD dengue Serotype 3; Pre-Injection 1 | 6.24 [5.57 to 6.99] | 5.95 [5.04 to 7.02]
  CYD dengue Serotype 3; Post-Injection 3: number analyzed (Participants) | 144 | 44
  CYD dengue Serotype 3; Post-Injection 3 | 136 [114 to 162] | 6.54 [5.20 to 8.22]
  CYD dengue Serotype 3; 1st year follow up: number analyzed (Participants) | 141 | 44
  CYD dengue Serotype 3; 1st year follow up | 25.4 [20.1 to 32.1] | 5.87 [5.00 to 6.89]
  CYD dengue Serotype 3; 2nd year follow up: number analyzed (Participants) | 133 | 41
  CYD dengue Serotype 3; 2nd year follow up | 29.9 [23.4 to 38.1] | 10.1 [6.68 to 15.20]
  CYD dengue Serotype 3; 3rd year follow up: number analyzed (Participants) | 134 | 43
  CYD dengue Serotype 3; 3rd year follow up | 14.6 [11.7 to 18.3] | 5.43 [4.83 to 6.10]
  CYD dengue Serotype 3; 4th year follow up: number analyzed (Participants) | 130 | 42
  CYD dengue Serotype 3; 4th year follow up | 11.4 [9.22 to 14.10] | 5.09 [4.91 to 5.29]
  CYD dengue Serotype 4; Pre-Injection 1: number analyzed (Participants) | 148 | 50
  CYD dengue Serotype 4; Pre-Injection 1 | 5.64 [5.20 to 6.11] | 5.39 [4.92 to 5.91]
  CYD dengue Serotype 4; Post-Injection 3: number analyzed (Participants) | 143 | 44
  CYD dengue Serotype 4; Post-Injection 3 | 104 [87.2 to 125] | 7.20 [5.74 to 9.05]
  CYD dengue Serotype 4; 1st year follow up: number analyzed (Participants) | 141 | 43
  CYD dengue Serotype 4; 1st year follow up | 31.8 [25.6 to 39.6] | 5.69 [4.70 to 6.89]
  CYD dengue Serotype 4; 2nd year follow up: number analyzed (Participants) | 140 | 43
  CYD dengue Serotype 4; 2nd year follow up | 30.6 [24.2 to 38.6] | 5.68 [4.74 to 6.82]
  CYD dengue Serotype 4; 3rd year follow up: number analyzed (Participants) | 132 | 43
  CYD dengue Serotype 4; 3rd year follow up | 22.3 [17.5 to 28.5] | 6.31 [4.84 to 8.24]
  CYD dengue Serotype 4; 4th year follow up: number analyzed (Participants) | 136 | 42
  CYD dengue Serotype 4; 4th year follow up | 16.5 [13.1 to 20.7] | 5.00 [5.00 to 5.00]

15. Secondary Outcome: GMTs of Antibodies in Participants 12 to 17 Years Old Against Each Serotype With the Parental Dengue Virus Strain Before and Following the Third Vaccination With CYD Dengue Vaccine or Placebo
Description: GMTs against each serotype with the dengue virus strain (parental strains) were assessed using a dengue PRNT assay.
Time Frame: as for outcome 8
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dilution)
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 141 | 46
Titers (1/dilution)
  CYD dengue Serotype 1; Pre-Injection 1 | 6.47 [5.31 to 7.89] | 5.47 [4.80 to 6.24]
  CYD dengue Serotype 1; Post-Injection 3: number analyzed (Participants) | 135 | 43
  CYD dengue Serotype 1; Post-Injection 3 | 28.5 [21.4 to 37.9] | 6.36 [5.12 to 7.89]
  CYD dengue Serotype 1; 1st year follow up: number analyzed (Participants) | 132 | 41
  CYD dengue Serotype 1; 1st year follow up | 9.69 [7.53 to 12.5] | 5.69 [4.88 to 6.63]
  CYD dengue Serotype 1; 2nd year follow up: number analyzed (Participants) | 128 | 40
  CYD dengue Serotype 1; 2nd year follow up | 8.31 [6.58 to 10.5] | 5.91 [4.80 to 7.27]
  CYD dengue Serotype 1; 3rd year follow up: number analyzed (Participants) | 124 | 40
  CYD dengue Serotype 1; 3rd year follow up | 8.02 [6.30 to 10.2] | 5.54 [4.79 to 6.39]
  CYD dengue Serotype 1; 4th year follow up: number analyzed (Participants) | 118 | 37
  CYD dengue Serotype 1; 4th year follow up | 7.41 [5.85 to 9.38] | 5.51 [4.80 to 6.34]
  CYD dengue Serotype 2; Pre-Injection 1 | 7.45 [5.95 to 9.33] | 5.54 [4.69 to 6.56]
  CYD dengue Serotype 2; Post-Injection 3: number analyzed (Participants) | 135 | 43
  CYD dengue Serotype 2; Post-Injection 3 | 48.7 [37.4 to 63.5] | 6.17 [5.03 to 7.58]
  CYD dengue Serotype 2; 1st year follow up: number analyzed (Participants) | 131 | 41
  CYD dengue Serotype 2; 1st year follow up | 16.6 [12.4 to 22.1] | 5.58 [4.78 to 6.52]
  CYD dengue Serotype 2; 2nd year follow up: number analyzed (Participants) | 128 | 40
  CYD dengue Serotype 2; 2nd year follow up | 18.7 [14.1 to 24.7] | 6.38 [4.92 to 8.27]
  CYD dengue Serotype 2; 3rd year follow up: number analyzed (Participants) | 124 | 40
  CYD dengue Serotype 2; 3rd year follow up | 13.3 [10.1 to 17.6] | 5.77 [4.71 to 7.07]
  CYD dengue Serotype 2; 4th year follow up: number analyzed (Participants) | 116 | 37
  CYD dengue Serotype 2; 4th year follow up | 14.0 [10.4 to 18.8] | 5.80 [4.68 to 7.17]
  CYD dengue Serotype 3; Pre-Injection 1: number analyzed (Participants) | 140 | 46
  CYD dengue Serotype 3; Pre-Injection 1 | 6.84 [5.81 to 8.06] | 6.83 [4.84 to 9.65]
  CYD dengue Serotype 3; Post-Injection 3: number analyzed (Participants) | 134 | 43
  CYD dengue Serotype 3; Post-Injection 3 | 71.4 [56.3 to 90.7] | 8.10 [5.66 to 11.6]
  CYD dengue Serotype 3; 1st year follow up: number analyzed (Participants) | 133 | 40
  CYD dengue Serotype 3; 1st year follow up | 19.7 [15.1 to 25.6] | 6.27 [4.55 to 8.64]
  CYD dengue Serotype 3; 2nd year follow up: number analyzed (Participants) | 126 | 40
  CYD dengue Serotype 3; 2nd year follow up | 20.5 [15.6 to 27.1] | 7.54 [5.16 to 11.0]
  CYD dengue Serotype 3; 3rd year follow up: number analyzed (Participants) | 123 | 40
  CYD dengue Serotype 3; 3rd year follow up | 15.3 [11.8 to 19.9] | 6.17 [4.58 to 8.31]
  CYD dengue Serotype 3; 4th year follow up: number analyzed (Participants) | 118 | 37
  CYD dengue Serotype 3; 4th year follow up | 13.7 [10.7 to 17.6] | 6.47 [4.49 to 9.30]
  CYD dengue Serotype 4; Pre-Injection 1: number analyzed (Participants) | 140 | 46
  CYD dengue Serotype 4; Pre-Injection 1 | 5.83 [5.17 to 6.56] | 5.08 [4.92 to 5.23]
  CYD dengue Serotype 4; Post-Injection 3: number analyzed (Participants) | 135 | 43
  CYD dengue Serotype 4; Post-Injection 3 | 79.2 [64.2 to 97.8] | 6.45 [4.89 to 8.53]
  CYD dengue Serotype 4; 1st year follow up: number analyzed (Participants) | 132 | 41
  CYD dengue Serotype 4; 1st year follow up | 30.8 [24.3 to 39] | 5.17 [4.84 to 5.52]
  CYD dengue Serotype 4; 2nd year follow up: number analyzed (Participants) | 128 | 40
  CYD dengue Serotype 4; 2nd year follow up | 33.4 [25.6 to 43.6] | 6.18 [4.99 to 7.65]
  CYD dengue Serotype 4; 3rd year follow up: number analyzed (Participants) | 123 | 40
  CYD dengue Serotype 4; 3rd year follow up | 23.1 [18.3 to 29.2] | 5.55 [4.79 to 6.42]
  CYD dengue Serotype 4; 4th year follow up: number analyzed (Participants) | 118 | 37
  CYD dengue Serotype 4; 4th year follow up | 20.8 [16.2 to 26.6] | 5.43 [4.92 to 6.00]

16. Secondary Outcome: GMTs of Antibodies in Participants 18 to 45 Years Old Against Each Serotype With the Parental Dengue Virus Strain Before and Following the Third Vaccination With CYD Dengue Vaccine or Placebo
Description: GMTs against each serotype with the dengue virus strain were assessed using a dengue PRNT assay.
Time Frame: as for outcome 8
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dilution)
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 521 | 174
Titers (1/dilution)
  CYD dengue Serotype 1; Pre-Injection 1: number analyzed (Participants) | 142 | 49
  CYD dengue Serotype 1; Pre-Injection 1 | 15.8 [11.7 to 21.5] | 19.2 [10.9 to 33.9]
  CYD dengue Serotype 1; Post-Injection 3: number analyzed (Participants) | 127 | 43
  CYD dengue Serotype 1; Post-Injection 3 | 48.7 [33.6 to 70.4] | 16.2 [9.77 to 27.0]
  CYD dengue Serotype 1; 1st year follow up: number analyzed (Participants) | 122 | 44
  CYD dengue Serotype 1; 1st year follow up | 26.3 [17.9 to 38.6] | 15.2 [8.76 to 26.3]
  CYD dengue Serotype 1; 2nd year follow up: number analyzed (Participants) | 117 | 41
  CYD dengue Serotype 1; 2nd year follow up | 26.3 [17.7 to 38.9] | 16.3 [9.09 to 29.3]
  CYD dengue Serotype 1; 3rd year follow up: number analyzed (Participants) | 114 | 39
  CYD dengue Serotype 1; 3rd year follow up | 24.1 [15.9 to 36.5] | 13.9 [7.89 to 24.6]
  CYD dengue Serotype 1; 4th year follow up: number analyzed (Participants) | 106 | 38
  CYD dengue Serotype 1; 4th year follow up | 23.5 [15.5 to 35.5] | 14.4 [8.03 to 25.6]
  CYD dengue Serotype 2; Pre-Injection 1: number analyzed (Participants) | 141 | 49
  CYD dengue Serotype 2; Pre-Injection 1 | 16.9 [12.3 to 23.1] | 21.0 [11.5 to 38.2]
  CYD dengue Serotype 2; Post-Injection 3: number analyzed (Participants) | 127 | 43
  CYD dengue Serotype 2; Post-Injection 3 | 66.9 [47.9 to 93.5] | 15.2 [8.61 to 27.0]
  CYD dengue Serotype 2; 1st year follow up: number analyzed (Participants) | 122 | 44
  CYD dengue Serotype 2; 1st year follow up | 50.4 [34.5 to 73.7] | 19.3 [10.7 to 34.7]
  CYD dengue Serotype 2; 2nd year follow up: number analyzed (Participants) | 117 | 41
  CYD dengue Serotype 2; 2nd year follow up | 66.5 [43.7 to 101] | 20.0 [10.2 to 39.0]
  CYD dengue Serotype 2; 3rd year follow up: number analyzed (Participants) | 114 | 39
  CYD dengue Serotype 2; 3rd year follow up | 38.4 [25.8 to 57.2] | 17.0 [9.38 to 30.8]
  CYD dengue Serotype 2; 4th year follow up: number analyzed (Participants) | 105 | 38
  CYD dengue Serotype 2; 4th year follow up | 32.9 [22.4 to 48.2] | 15.5 [8.51 to 28.2]
  CYD dengue Serotype 3; Pre-Injection 1: number analyzed (Participants) | 141 | 48
  CYD dengue Serotype 3; Pre-Injection 1 | 14.5 [11.2 to 18.7] | 19.4 [11.4 to 33.1]
  CYD dengue Serotype 3; Post-Injection 3: number analyzed (Participants) | 127 | 43
  CYD dengue Serotype 3; Post-Injection 3 | 88.4 [68.6 to 114] | 13.3 [8.22 to 21.7]
  CYD dengue Serotype 3; 1st year follow up: number analyzed (Participants) | 121 | 44
  CYD dengue Serotype 3; 1st year follow up | 45.2 [32.1 to 63.6] | 14.8 [8.96 to 24.3]
  CYD dengue Serotype 3; 2nd year follow up: number analyzed (Participants) | 117 | 41
  CYD dengue Serotype 3; 2nd year follow up | 64.8 [46.8 to 89.7] | 19.9 [11.5 to 34.5]
  CYD dengue Serotype 3; 3rd year follow up: number analyzed (Participants) | 112 | 39
  CYD dengue Serotype 3; 3rd year follow up | 48.3 [33.0 to 70.8] | 14.7 [8.46 to 25.7]
  CYD dengue Serotype 3; 4th year follow up: number analyzed (Participants) | 106 | 37
  CYD dengue Serotype 3; 4th year follow up | 28.6 [20.2 to 40.6] | 11.8 [7.18 to 19.3]
  CYD dengue Serotype 4; Pre-Injection 1: number analyzed (Participants) | 140 | 48
  CYD dengue Serotype 4; Pre-Injection 1 | 10.1 [8.03 to 12.7] | 11.7 [7.74 to 17.6]
  CYD dengue Serotype 4; Post-Injection 3: number analyzed (Participants) | 126 | 43
  CYD dengue Serotype 4; Post-Injection 3 | 122 [96.5 to 155] | 10.0 [6.96 to 14.4]
  CYD dengue Serotype 4; 1st year follow up: number analyzed (Participants) | 122 | 44
  CYD dengue Serotype 4; 1st year follow up | 70.3 [53.6 to 92.2] | 9.87 [6.88 to 14.2]
  CYD dengue Serotype 4; 2nd year follow up: number analyzed (Participants) | 117 | 41
  CYD dengue Serotype 4; 2nd year follow up | 52.6 [39.9 to 69.3] | 8.50 [6.07 to 11.9]
  CYD dengue Serotype 4; 3rd year follow up: number analyzed (Participants) | 114 | 39
  CYD dengue Serotype 4; 3rd year follow up | 46.4 [35.5 to 60.6] | 8.39 [5.83 to 12.1]
  CYD dengue Serotype 4; 4th year follow up: number analyzed (Participants) | 107 | 38
  CYD dengue Serotype 4; 4th year follow up | 32.6 [25.2 to 42.3] | 7.54 [5.69 to 10.0]

17. Secondary Outcome: Percentage of Participants (Aged 2 to 11 Years) Immune to Dengue at Baseline Who Are Seropositive for Each of the Dengue Virus Serotypes up to 4 Years After the Third Vaccination With CYD Dengue Vaccine or Placebo
Description: Seropositivity against each serotype with the dengue virus strain were assessed using a dengue PRNT assay. Seropositive participants were defined as participants with antibody titers >=10 (1/dilution). Dengue participants immune at baseline was defined as those participants with titers >=10 (1/dilution) against at least one dengue serotype at baseline.
Time Frame: 28 days Post-Injection 3, at 1 year follow up, 2 year follow up, 3 year follow up and 4 year follow up (assessed post-injection 3 during the follow up duration of 4 years)
Population: as for outcome 9
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 29 | 13
Percentage of participants
  CYD dengue Serotype 1; Post-Injection 3: number analyzed (Participants) | 27 | 13
  CYD dengue Serotype 1; Post-Injection 3 | 96.3 | 0.0
  CYD dengue Serotype 1; 1st year follow up: number analyzed (Participants) | 27 | 13
  CYD dengue Serotype 1; 1st year follow up | 74.1 | 7.7
  CYD dengue Serotype 1; 2nd year follow up: number analyzed (Participants) | 27 | 12
  CYD dengue Serotype 1; 2nd year follow up | 55.6 | 0.0
  CYD dengue Serotype 1; 3rd year follow up: number analyzed (Participants) | 27 | 12
  CYD dengue Serotype 1; 3rd year follow up | 33.3 | 0.0
  CYD dengue Serotype 1; 4th year follow up: number analyzed (Participants) | 27 | 12
  CYD dengue Serotype 1; 4th year follow up | 22.2 | 0.0
  CYD dengue Serotype 2; Post-Injection 3: number analyzed (Participants) | 27 | 13
  CYD dengue Serotype 2; Post-Injection 3 | 100.0 | 15.4
  CYD dengue Serotype 2; 1st year follow up: number analyzed (Participants) | 27 | 13
  CYD dengue Serotype 2; 1st year follow up | 85.2 | 15.4
  CYD dengue Serotype 2; 2nd year follow up: number analyzed (Participants) | 27 | 12
  CYD dengue Serotype 2; 2nd year follow up | 66.7 | 16.7
  CYD dengue Serotype 2; 3rd year follow up: number analyzed (Participants) | 27 | 12
  CYD dengue Serotype 2; 3rd year follow up | 48.1 | 16.7
  CYD dengue Serotype 2; 4th year follow up: number analyzed (Participants) | 27 | 12
  CYD dengue Serotype 2; 4th year follow up | 48.1 | 0.0
  CYD dengue Serotype 3; Post-Injection 3: number analyzed (Participants) | 27 | 13
  CYD dengue Serotype 3; Post-Injection 3 | 100.0 | 23.1
  CYD dengue Serotype 3; 1st year follow up: number analyzed (Participants) | 27 | 13
  CYD dengue Serotype 3; 1st year follow up | 88.9 | 7.7
  CYD dengue Serotype 3; 2nd year follow up: number analyzed (Participants) | 27 | 12
  CYD dengue Serotype 3; 2nd year follow up | 81.5 | 16.7
  CYD dengue Serotype 3; 3rd year follow up: number analyzed (Participants) | 27 | 12
  CYD dengue Serotype 3; 3rd year follow up | 59.3 | 8.3
  CYD dengue Serotype 3; 4th year follow up: number analyzed (Participants) | 24 | 12
  CYD dengue Serotype 3; 4th year follow up | 50.0 | 0.0
  CYD dengue Serotype 4; Post-Injection 3: number analyzed (Participants) | 26 | 13
  CYD dengue Serotype 4; Post-Injection 3 | 100.0 | 23.1
  CYD dengue Serotype 4; 1st year follow up: number analyzed (Participants) | 27 | 13
  CYD dengue Serotype 4; 1st year follow up | 88.9 | 15.4
  CYD dengue Serotype 4; 2nd year follow up: number analyzed (Participants) | 27 | 12
  CYD dengue Serotype 4; 2nd year follow up | 74.1 | 0.0
  CYD dengue Serotype 4; 3rd year follow up: number analyzed (Participants) | 27 | 12
  CYD dengue Serotype 4; 3rd year follow up | 70.4 | 16.7
  CYD dengue Serotype 4; 4th year follow up: number analyzed (Participants) | 27 | 12
  CYD dengue Serotype 4; 4th year follow up | 70.4 | 0.0

18. Secondary Outcome: Percentage of Participants (Aged 2 to 11 Years) Naïve to Dengue at Baseline Who Are Seropositive for Each of the Dengue Virus Serotypes up to 4 Years After the Third Vaccination With CYD Dengue Vaccine or Placebo
Description: Seropositivity against each serotype with the dengue virus strain were assessed using a dengue PRNT assay. Seropositive participants were defined as participants with neutralizing antibody titers >=10 (1/dilution). Dengue participants naïve at baseline was defined as those participants with titers <10 (1/dilution) against all dengue serotypes at baseline.
Time Frame: as for outcome 17
Population: as for outcome 9
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 118 | 37
Percentage of participants
  CYD dengue Serotype 1; Post-Injection 3: number analyzed (Participants) | 115 | 32
  CYD dengue Serotype 1; Post-Injection 3 | 89.6 | 12.5
  CYD dengue Serotype 1; 1st year follow up: number analyzed (Participants) | 113 | 31
  CYD dengue Serotype 1; 1st year follow up | 33.6 | 6.5
  CYD dengue Serotype 1; 2nd year follow up: number analyzed (Participants) | 112 | 31
  CYD dengue Serotype 1; 2nd year follow up | 20.5 | 0.0
  CYD dengue Serotype 1; 3rd year follow up: number analyzed (Participants) | 105 | 31
  CYD dengue Serotype 1; 3rd year follow up | 12.4 | 0.0
  CYD dengue Serotype 1; 4th year follow up: number analyzed (Participants) | 108 | 30
  CYD dengue Serotype 1; 4th year follow up | 6.5 | 0.0
  CYD dengue Serotype 2; Post-Injection 3: number analyzed (Participants) | 115 | 32
  CYD dengue Serotype 2; Post-Injection 3 | 93.0 | 12.5
  CYD dengue Serotype 2; 1st year follow up: number analyzed (Participants) | 113 | 32
  CYD dengue Serotype 2; 1st year follow up | 54.0 | 6.3
  CYD dengue Serotype 2; 2nd year follow up: number analyzed (Participants) | 112 | 31
  CYD dengue Serotype 2; 2nd year follow up | 49.1 | 9.7
  CYD dengue Serotype 2; 3rd year follow up: number analyzed (Participants) | 106 | 31
  CYD dengue Serotype 2; 3rd year follow up | 31.1 | 3.2
  CYD dengue Serotype 2; 4th year follow up: number analyzed (Participants) | 102 | 30
  CYD dengue Serotype 2; 4th year follow up | 34.3 | 3.3
  CYD dengue Serotype 3; Post-Injection 3: number analyzed (Participants) | 115 | 31
  CYD dengue Serotype 3; Post-Injection 3 | 97.4 | 9.7
  CYD dengue Serotype 3; 1st year follow up: number analyzed (Participants) | 113 | 31
  CYD dengue Serotype 3; 1st year follow up | 60.2 | 9.7
  CYD dengue Serotype 3; 2nd year follow up: number analyzed (Participants) | 105 | 29
  CYD dengue Serotype 3; 2nd year follow up | 72.4 | 34.5
  CYD dengue Serotype 3; 3rd year follow up: number analyzed (Participants) | 106 | 31
  CYD dengue Serotype 3; 3rd year follow up | 47.2 | 3.2
  CYD dengue Serotype 3; 4th year follow up: number analyzed (Participants) | 105 | 30
  CYD dengue Serotype 3; 4th year follow up | 34.3 | 3.3
  CYD dengue Serotype 4; Post-Injection 3: number analyzed (Participants) | 115 | 31
  CYD dengue Serotype 4; Post-Injection 3 | 96.5 | 19.4
  CYD dengue Serotype 4; 1st year follow: number analyzed (Participants) | 113 | 30
  CYD dengue Serotype 4; 1st year follow | 71.7 | 0.0
  CYD dengue Serotype 4; 2nd year follow up: number analyzed (Participants) | 112 | 31
  CYD dengue Serotype 4; 2nd year follow up | 73.2 | 6.5
  CYD dengue Serotype 4; 3rd year follow up: number analyzed (Participants) | 104 | 31
  CYD dengue Serotype 4; 3rd year follow up | 58.7 | 3.2
  CYD dengue Serotype 4; 4th year follow up: number analyzed (Participants) | 108 | 30
  CYD dengue Serotype 4; 4th year follow up | 44.4 | 0.0

19. Secondary Outcome: Percentage of Participants (Aged 12 to 17 Years) Immune to Dengue at Baseline Who Are Seropositive for Each of the Dengue Virus Serotypes up to 4 Years After the Third Vaccination With CYD Dengue Vaccine or Placebo
Description: Seropositivity against each serotype with the dengue virus strain were assessed using a dengue PRNT assay. Seropositive participants were defined as participants with neutralizing antibody titers >=10 (1/dilution). Dengue participants immune at baseline was defined as those participants with titers >=10 (1/dilution) against at least one dengue serotype at baseline.
Time Frame: as for outcome 17
Population: as for outcome 9
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 19 | 7
Percentage of participants
  CYD dengue Serotype 1; Post-Injection 3: number analyzed (Participants) | 18 | 6
  CYD dengue Serotype 1; Post-Injection 3 | 94.4 | 33.3
  CYD dengue Serotype 1; 1st year follow up: number analyzed (Participants) | 17 | 5
  CYD dengue Serotype 1; 1st year follow up | 58.8 | 20.0
  CYD dengue Serotype 1; 2nd year follow up: number analyzed (Participants) | 15 | 6
  CYD dengue Serotype 1; 2nd year follow up | 46.7 | 16.7
  CYD dengue Serotype 1; 3rd year follow up: number analyzed (Participants) | 16 | 6
  CYD dengue Serotype 1; 3rd year follow up | 43.8 | 16.7
  CYD dengue Serotype 1; 4th year follow up: number analyzed (Participants) | 14 | 5
  CYD dengue Serotype 1; 4th year follow up | 42.9 | 20.0
  CYD dengue Serotype 2; Post-Injection 3: number analyzed (Participants) | 18 | 6
  CYD dengue Serotype 2; Post-Injection 3 | 94.4 | 16.7
  CYD dengue Serotype 2; 1st year follow up: number analyzed (Participants) | 17 | 5
  CYD dengue Serotype 2; 1st year follow up | 82.4 | 20.0
  CYD dengue Serotype 2; 2nd year follow up: number analyzed (Participants) | 15 | 6
  CYD dengue Serotype 2; 2nd year follow up | 73.3 | 33.3
  CYD dengue Serotype 2; 3rd year follow up: number analyzed (Participants) | 16 | 6
  CYD dengue Serotype 2; 3rd year follow up | 68.8 | 16.7
  CYD dengue Serotype 2; 4th year follow up: number analyzed (Participants) | 14 | 5
  CYD dengue Serotype 2; 4th year follow up | 71.4 | 20.0
  CYD dengue Serotype 3; Post-Injection 3: number analyzed (Participants) | 18 | 6
  CYD dengue Serotype 3; Post-Injection 3 | 100.0 | 50.0
  CYD dengue Serotype 3; 1st year follow up: number analyzed (Participants) | 17 | 5
  CYD dengue Serotype 3; 1st year follow up | 76.5 | 20.0
  CYD dengue Serotype 3; 2nd year follow up: number analyzed (Participants) | 15 | 6
  CYD dengue Serotype 3; 2nd year follow up | 80.0 | 50.0
  CYD dengue Serotype 3; 3rd year follow up: number analyzed (Participants) | 16 | 6
  CYD dengue Serotype 3; 3rd year follow up | 68.8 | 16.7
  CYD dengue Serotype 3; 4th year follow up: number analyzed (Participants) | 14 | 5
  CYD dengue Serotype 3; 4th year follow up | 71.4 | 20.0
  CYD dengue Serotype 4; Post-Injection 3: number analyzed (Participants) | 18 | 6
  CYD dengue Serotype 4; Post-Injection 3 | 100.0 | 33.3
  CYD dengue Serotype 4; 1st year follow up: number analyzed (Participants) | 17 | 5
  CYD dengue Serotype 4; 1st year follow up | 100.0 | 20.0
  CYD dengue Serotype 4; 2nd year follow up: number analyzed (Participants) | 15 | 6
  CYD dengue Serotype 4; 2nd year follow up | 100.0 | 16.7
  CYD dengue Serotype 4; 3rd year follow up: number analyzed (Participants) | 16 | 6
  CYD dengue Serotype 4; 3rd year follow up | 93.8 | 16.7
  CYD dengue Serotype 4; 4th year follow up: number analyzed (Participants) | 14 | 5
  CYD dengue Serotype 4; 4th year follow up | 100.0 | 20.0

20. Secondary Outcome: Percentage of Participants (Aged 12 to 17 Years) Naïve to Dengue at Baseline Who Are Seropositive for Each of the Dengue Virus Serotypes up to 4 Years After the Third Vaccination With CYD Dengue Vaccine or Placebo
Description: Seropositivity against each serotype with the dengue virus strain were assessed using a PRNT assay. Seropositive participants were defined as participants with neutralizing antibody titers >=10 (1/dilution). Dengue participants naïve at baseline was defined as those participants with titers <10 (1/dilution) against all dengue serotypes at baseline.
Time Frame: as for outcome 17
Population: as for outcome 9
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 121 | 39
Percentage of participants
  CYD dengue Serotype 1; Post-Injection 3: number analyzed (Participants) | 116 | 37
  CYD dengue Serotype 1; Post-Injection 3 | 62.9 | 8.1
  CYD dengue Serotype 1; 1st year follow up: number analyzed (Participants) | 115 | 36
  CYD dengue Serotype 1; 1st year follow up | 20.9 | 5.6
  CYD dengue Serotype 1; 2nd year follow up: number analyzed (Participants) | 112 | 34
  CYD dengue Serotype 1; 2nd year follow up | 16.1 | 5.9
  CYD dengue Serotype 1; 3rd year follow up: number analyzed (Participants) | 108 | 34
  CYD dengue Serotype 1; 3rd year follow up | 12.0 | 2.9
  CYD dengue Serotype 1; 4th year follow up: number analyzed (Participants) | 104 | 32
  CYD dengue Serotype 1; 4th year follow up | 7.7 | 3.1
  CYD dengue Serotype 2; Post-Injection 3: number analyzed (Participants) | 116 | 37
  CYD dengue Serotype 2; Post-Injection 3 | 81.9 | 8.1
  CYD dengue Serotype 2; 1st year follow up: number analyzed (Participants) | 114 | 36
  CYD dengue Serotype 2; 1st year follow up | 38.6 | 2.8
  CYD dengue Serotype 2; 2nd year follow up: number analyzed (Participants) | 112 | 34
  CYD dengue Serotype 2; 2nd year follow up | 49.1 | 5.9
  CYD dengue Serotype 2; 3rd year follow up: number analyzed (Participants) | 108 | 34
  CYD dengue Serotype 2; 3rd year follow up | 30.6 | 2.9
  CYD dengue Serotype 2; 4th year follow up: number analyzed (Participants) | 102 | 32
  CYD dengue Serotype 2; 4th year follow up | 31.4 | 3.1
  CYD dengue Serotype 3; Post-Injection 3: number analyzed (Participants) | 115 | 37
  CYD dengue Serotype 3; Post-Injection 3 | 87.0 | 16.2
  CYD dengue Serotype 3; 1st year follow up: number analyzed (Participants) | 116 | 35
  CYD dengue Serotype 3; 1st year follow up | 59.5 | 2.9
  CYD dengue Serotype 3; 2nd year follow up: number analyzed (Participants) | 110 | 34
  CYD dengue Serotype 3; 2nd year follow up | 53.6 | 5.9
  CYD dengue Serotype 3; 3rd year follow up: number analyzed (Participants) | 107 | 34
  CYD dengue Serotype 3; 3rd year follow up | 45.8 | 2.9
  CYD dengue Serotype 3; 4th year follow up: number analyzed (Participants) | 104 | 32
  CYD dengue Serotype 3; 4th year follow up | 44.2 | 3.1
  CYD dengue Serotype 4; Post-Injection 3: number analyzed (Participants) | 116 | 37
  CYD dengue Serotype 4; Post-Injection 3 | 89.7 | 5.4
  CYD dengue Serotype 4; 1st year follow up: number analyzed (Participants) | 115 | 36
  CYD dengue Serotype 4; 1st year follow up | 69.6 | 0.0
  CYD dengue Serotype 4; 2nd year follow up: number analyzed (Participants) | 112 | 34
  CYD dengue Serotype 4; 2nd year follow up | 67.0 | 8.8
  CYD dengue Serotype 4; 3rd year follow up: number analyzed (Participants) | 107 | 34
  CYD dengue Serotype 4; 3rd year follow up | 62.6 | 2.9
  CYD dengue Serotype 4; 4th year follow up: number analyzed (Participants) | 104 | 32
  CYD dengue Serotype 4; 4th year follow up | 55.8 | 6.3

21. Secondary Outcome: Percentage of Participants (Aged 18 to 45 Years) Immune to Dengue at Baseline Who Are Seropositive for Each of the Dengue Virus Serotypes up to 4 Years After the Third Vaccination With CYD Dengue Vaccine or Placebo
Description: as for outcome 19
Time Frame: as for outcome 17
Population: as for outcome 9
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 66 | 27
Percentage of participants
  CYD dengue Serotype 1; Post-Injection 3: number analyzed (Participants) | 56 | 20
  CYD dengue Serotype 1; Post-Injection 3 | 89.3 | 70.0
  CYD dengue Serotype 1; 1st year follow up: number analyzed (Participants) | 54 | 21
  CYD dengue Serotype 1; 1st year follow up | 77.8 | 57.1
  CYD dengue Serotype 1; 2nd year follow up: number analyzed (Participants) | 51 | 20
  CYD dengue Serotype 1; 2nd year follow up | 86.3 | 65.0
  CYD dengue Serotype 1; 3rd year follow up: number analyzed (Participants) | 52 | 19
  CYD dengue Serotype 1; 3rd year follow up | 80.8 | 63.2
  CYD dengue Serotype 1; 4th year follow up: number analyzed (Participants) | 46 | 18
  CYD dengue Serotype 1; 4th year follow up | 84.8 | 66.7
  CYD dengue Serotype 2; Post-Injection 3: number analyzed (Participants) | 56 | 20
  CYD dengue Serotype 2; Post-Injection 3 | 91.1 | 65.0
  CYD dengue Serotype 2; 1st year follow up: number analyzed (Participants) | 54 | 21
  CYD dengue Serotype 2; 1st year follow up | 88.9 | 71.4
  CYD dengue Serotype 2; 2nd year follow up: number analyzed (Participants) | 51 | 20
  CYD dengue Serotype 2; 2nd year follow up | 92.2 | 70.0
  CYD dengue Serotype 2; 3rd year follow up: number analyzed (Participants) | 52 | 19
  CYD dengue Serotype 2; 3rd year follow up | 88.5 | 68.4
  CYD dengue Serotype 2; 4th year follow up: number analyzed (Participants) | 47 | 18
  CYD dengue Serotype 2; 4th year follow up | 91.5 | 66.7
  CYD dengue Serotype 3; Post-Injection 3: number analyzed (Participants) | 56 | 20
  CYD dengue Serotype 3; Post-Injection 3 | 98.2 | 60.0
  CYD dengue Serotype 3; 1st year follow up: number analyzed (Participants) | 54 | 21
  CYD dengue Serotype 3; 1st year follow up | 90.7 | 66.7
  CYD dengue Serotype 3; 2nd year follow up: number analyzed (Participants) | 51 | 20
  CYD dengue Serotype 3; 2nd year follow up | 98.0 | 70.0
  CYD dengue Serotype 3; 3rd year follow up: number analyzed (Participants) | 52 | 19
  CYD dengue Serotype 3; 3rd year follow up | 94.2 | 73.7
  CYD dengue Serotype 3; 4th year follow up: number analyzed (Participants) | 47 | 18
  CYD dengue Serotype 3; 4th year follow up | 91.5 | 61.1
  CYD dengue Serotype 4; Post-Injection 3: number analyzed (Participants) | 55 | 20
  CYD dengue Serotype 4; Post-Injection 3 | 100.0 | 65.0
  CYD dengue Serotype 4; 1st year follow up: number analyzed (Participants) | 54 | 21
  CYD dengue Serotype 4; 1st year follow up | 98.1 | 47.6
  CYD dengue Serotype 4; 2nd year follow up: number analyzed (Participants) | 51 | 20
  CYD dengue Serotype 4; 2nd year follow up | 96.1 | 45.0
  CYD dengue Serotype 4; 3rd year follow up: number analyzed (Participants) | 52 | 19
  CYD dengue Serotype 4; 3rd year follow up | 100.0 | 42.1
  CYD dengue Serotype 4; 4th year follow up: number analyzed (Participants) | 47 | 18
  CYD dengue Serotype 4; 4th year follow up | 97.9 | 44.4

22. Secondary Outcome: Percentage of Participants (Aged 18 to 45 Years) Naïve to Dengue at Baseline Who Are Seropositive for Each of the Dengue Virus Serotypes up to 4 Years After the Third Vaccination With CYD Dengue Vaccine or Placebo
Description: as for outcome 18
Time Frame: as for outcome 17
Population: as for outcome 9
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 74 | 22
Percentage of participants
  CYD dengue Serotype 1; Post-Injection 3: number analyzed (Participants) | 64 | 21
  CYD dengue Serotype 1; Post-Injection 3 | 59.4 | 14.3
  CYD dengue Serotype 1; 1st year follow up: number analyzed (Participants) | 61 | 21
  CYD dengue Serotype 1; 1st year follow up | 21.3 | 9.5
  CYD dengue Serotype 1; 2nd year follow up: number analyzed (Participants) | 59 | 19
  CYD dengue Serotype 1; 2nd year follow up | 10.2 | 5.3
  CYD dengue Serotype 1; 3rd year follow up: number analyzed (Participants) | 56 | 18
  CYD dengue Serotype 1; 3rd year follow up | 7.1 | 0
  CYD dengue Serotype 1; 4th year follow up: number analyzed (Participants) | 54 | 18
  CYD dengue Serotype 1; 4th year follow up | 5.6 | 0
  CYD dengue Serotype 2; Post-Injection 3: number analyzed (Participants) | 64 | 21
  CYD dengue Serotype 2; Post-Injection 3 | 73.4 | 0
  CYD dengue Serotype 2; 1st year follow up: number analyzed (Participants) | 61 | 21
  CYD dengue Serotype 2; 1st year follow up | 49.2 | 14.3
  CYD dengue Serotype 2; 2nd year follow up: number analyzed (Participants) | 59 | 19
  CYD dengue Serotype 2; 2nd year follow up | 50.8 | 0
  CYD dengue Serotype 2; 3rd year follow up: number analyzed (Participants) | 56 | 18
  CYD dengue Serotype 2; 3rd year follow up | 28.6 | 5.6
  CYD dengue Serotype 2; 4th year follow up: number analyzed (Participants) | 53 | 18
  CYD dengue Serotype 2; 4th year follow up | 26.4 | 0
  CYD dengue Serotype 3; Post-Injection 3: number analyzed (Participants) | 64 | 21
  CYD dengue Serotype 3; Post-Injection 3 | 87.5 | 14.3
  CYD dengue Serotype 3; 1st year follow up: number analyzed (Participants) | 60 | 21
  CYD dengue Serotype 3; 1st year follow up | 48.3 | 14.3
  CYD dengue Serotype 3; 2nd year follow up: number analyzed (Participants) | 59 | 19
  CYD dengue Serotype 3; 2nd year follow up | 61.0 | 21.1
  CYD dengue Serotype 3; 3rd year follow up: number analyzed (Participants) | 54 | 18
  CYD dengue Serotype 3; 3rd year follow up | 46.3 | 0
  CYD dengue Serotype 3; 4th year follow up: number analyzed (Participants) | 53 | 17
  CYD dengue Serotype 3; 4th year follow up | 28.3 | 0
  CYD dengue Serotype 4; Post-Injection 3: number analyzed (Participants) | 64 | 21
  CYD dengue Serotype 4; Post-Injection 3 | 87.5 | 4.8
  CYD dengue Serotype 4; 1st year follow up: number analyzed (Participants) | 61 | 21
  CYD dengue Serotype 4; 1st year follow up | 78.7 | 14.3
  CYD dengue Serotype 4; 2nd year follow up: number analyzed (Participants) | 59 | 19
  CYD dengue Serotype 4; 2nd year follow up | 71.2 | 5.3
  CYD dengue Serotype 4; 3rd year follow up: number analyzed (Participants) | 56 | 18
  CYD dengue Serotype 4; 3rd year follow up | 66.1 | 0
  CYD dengue Serotype 4; 4th year follow up: number analyzed (Participants) | 54 | 18
  CYD dengue Serotype 4; 4th year follow up | 63.0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AE) were collected from Day 0 (post-vaccination) up to the end of 4th year of follow up (up to 60 months).
Description: Solicited reaction (SR) was an adverse reaction observed and reported under conditions (nature and onset) prelisted (i.e., solicited) in the electronic case report form (eCRF). An unsolicited AE was an observed AE that did not fulfill conditions prelisted in eCRF in terms of symptom and/or onset post-vaccination. Safety analysis set.
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 3/898 | 0/300
Serious Adverse Events (participants affected / at risk) | 43/898 | 13/300
Other Adverse Events (participants affected / at risk) | 481/898 | 198/300
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CYD Dengue Vaccine Group (N=898) | Placebo Group (N=300)
Osteotomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Ruptured ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Adverse drug reaction (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 2 (2) | 0 (0)
Radial nerve palsy (Nervous system disorders) | 1 (1) | 0 (0)
Syncope vasovagal (Nervous system disorders) | 1 (1) | 0 (0)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingivitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Thyroid disorder (Endocrine disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis viral (Infections and infestations) | 2 (2) | 0 (0)
Corneal infection (Infections and infestations) | 1 (1) | 0 (0)
Dengue fever (Infections and infestations) | 3 (3) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (3) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 2 (2)
Groin abscess (Infections and infestations) | 1 (1) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 2 (2) | 0 (0)
Herpangina (Infections and infestations) | 1 (1) | 0 (0)
Lymph node tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Meningitis viral (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Pharyngitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | CYD Dengue Vaccine Group (N=898) | Placebo Group (N=300)
Cough (Respiratory, thoracic and mediastinal disorders) | 42 (48) | 15 (17)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 42 (47) | 15 (15)
Headache; Post-Any Injection (Nervous system disorders) | 402/891 (402) | 114/297 (114)
Injection site Pain; Post-Any Injection (General disorders) | 481/892 (481) | 198/297 (198)
Injection site Erythema; Post-Any Injection (General disorders) | 64/891 (64) | 45/297 (45)
Injection site Swelling; Post-Any Injection (General disorders) | 37/892 (37) | 25/297 (25)
Fever; Post-Any Injection (General disorders) | 101/892 (101) | 22/297 (22)
Malaise; Post-Any Injection (General disorders) | 372/891 (372) | 105/297 (105)
Asthenia; Post-Any Injection (General disorders) | 183/891 (183) | 52/297 (52)
Myalgia; Post-Any Injection (Musculoskeletal and connective tissue disorders) | 394/891 (394) | 130/297 (130)
Upper respiratory tract infection (Infections and infestations) | 72 (77) | 27 (30)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.